# I3Y-MC-JPBK

I3Y-MC-JPBK: A Randomized Phase 3 Study of Abemaciclib plus Best Supportive Care versus Erlotinib plus Best Supportive Care in Patients with Stage IV NSCLC with a Detectable *KRAS* Mutation Who Have Progressed After Platinum-Based Chemotherapy

NCT02152631

Approval Date: May 13, 2014

# 1. Protocol I3Y-MC-JPBK A Randomized Phase 3 Study of LY2835219 plus Best Supportive Care versus Erlotinib plus Best Supportive Care in Patients with Stage IV NSCLC with a Detectable KRAS Mutation Who Have Progressed After Platinum-Based Chemotherapy

### **Confidential Information**

The information contained in this protocol is confidential and is intended for the use of clinical investigators. It is the property of Eli Lilly and Company or its subsidiaries and should not be copied by or distributed to persons not involved in the clinical investigation of LY2835219, unless such persons are bound by a confidentiality agreement with Eli Lilly and Company or its subsidiaries. This document and its associated attachments are subject to United States Freedom of Information Act Exemption 4.

### LY2835219

This study is a global, multicenter, randomized, open-label, Phase 3 trial in patients with Stage IV NSCLC whose tumors have a detectable *KRAS* mutation in codons 12 or 13 and who have progressed after platinum-based chemotherapy and received 1 other prior therapy or are ineligible for further chemotherapy randomized to receive either LY2835219 plus best supportive care or erlotinib plus best supportive care.

Eli Lilly and Company Indianapolis, Indiana USA 46285

Protocol Electronically Signed and Approved by Lilly on date provided below.

Approval Date: 13-May-2014 GMT

# 2. Synopsis

### **Study Rationale**

Patients with metastatic non-small cell lung cancer (NSCLC) that harbor *KRAS* mutations (25%) have a poor prognosis compared to NSCLC patients who are *KRAS* wild-type. The p16INK4A-cyclin D-cyclin-dependent kinases (CDK) 4/6-retinoblastoma pathway is frequently dysregulated in NSCLC and therefore this pathway represents an attractive therapeutic target. LY2835219 is a potent and selective small molecule inhibitor of CDK4/6 that has shown acceptable safety/tolerability as well as evidence of clinical activity in multiple tumor types.

The Phase 3 Study I3Y-MC-JPBK (JPBK) study will evaluate the clinical activity of LY2835219 plus best supportive care (BSC) versus erlotinib plus BSC for patients with Stage IV NSCLC whose tumors have a detectable *KRAS* mutation (specifically, in codons 12 or 13 of the *KRAS* oncogene as determined by an investigational assay at the Study JPBK central laboratory) and who have progressed after prior platinum-based therapy and received 1 other prior therapy or are not eligible for further chemotherapy.

### Clinical Protocol Synopsis: Study I3Y-MC-JPBK

| Name of Investigational Product: LY2835219 |
|---|
| <b>Title of Study:</b> A randomized Phase 3 study of LY2835219 plus best supportive care versus erlotinib plus best |
| supportive care in patients with Stage IV NSCLC with a detectable KRAS mutation who have progressed after |
| platinum-based chemotherapy. |
| Number of Planned Patients: Phase of Development: 3 |
| Entered: 2500 |
| Enrolled/Randomized: 550 |
| Completed: 550 |
| T (1 CC) 1 A : (1 CA (1 |

**Length of Study:** Approximately 34 months Planned first patient visit: September 2014

Planned last patient visit: excluding the extension period: July 2017

Planned interim analysis: Analysis for safety will occur every 6 months. One futility analysis will occur after

100 progression-free survival (PFS) events have been observed.

**Objectives:** The co-primary objectives of this study are to compare LY2835219 plus BSC versus erlotinib plus BSC in patients with Stage IV NSCLC whose tumors have detectable *KRAS* mutations (specifically, in codons 12 or 13 of the *KRAS* oncogene as determined by an investigational assay at the Study JPBK central laboratory) and who have progressed after prior platinum-based therapy and 1 other prior therapy or are not eligible for further chemotherapy with respect to:

- PFS
- overall survival (OS)

The secondary objectives of the study are to compare LY2835219 plus BSC to erlotinib plus BSC with respect to:

- overall response rate (complete response + partial response)
- changes in patient-reported pain and disease-related symptoms collected via the MD Anderson Symptom Inventory (MDASI-LC) and changes in health status via European Quality of Life – 5 Dimensions – 5 Level (EQ-5D 5L)
- safety and tolerability
- resource utilization (for example, analgesic type, hospitalization, transfusion)
- the pharmacokinetic (PK)/pharmacodynamic properties of LY2835219

The exploratory objectives of the study are as follows:

 to explore biomarkers relevant to LY2835219 and the disease state and to correlate these markers to clinical outcome and to LY2835219

**Study Design:** Study I3Y-MC-JPBK is a multicenter, randomized, open-label, parallel, comparator-controlled trial in patients with Stage IV NSCLC whose tumors have a detectable *KRAS* mutation in codons 12 or 13 by an investigational assay and who have progressed after platinum-based chemotherapy and received 1 other prior therapy or are ineligible for further chemotherapy after platinum-based therapy.

Diagnosis and Main Criteria for Inclusion and Exclusions: Patients will be males or females who are ≥18 years of age with a confirmed diagnosis of stage IV NSCLC according to American Joint Committee on Cancer Staging Handbook 7th edition. The patient's tumor will have a mutation in codon 12 or 13 of the *KRAS* oncogene, and the patient must have progressed after platinum-based chemotherapy (with or without maintenance therapy) AND has received 1 other prior chemotherapy for advanced and/or metastatic disease OR is judged by the physician as ineligible for further standard second-line chemotherapy. Patients may not have received prior epidermal growth factor receptor (EGFR)-targeted therapy, including any multitarget tyrosine kinase inhibitors, which may inhibit EGFR. Patients will have measureable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1), adequate tumor-derived material from biopsy or surgery for analysis of *KRAS* status, an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1, and adequate organ function. Patients will be excluded from the study if they have a personal history of certain heart disease, presence of unstable central nervous system metastasis, or history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix) unless in complete remission with no therapy for a minimum of 3 years.

**Test Product, Dosage, and Mode of Administration:** LY2835219 200 mg administered orally as capsules every 12 hours

### **Planned Duration of Treatment:**

Treatment period: until disease progression or unacceptable toxicity occurs (or both)

Short-term follow-up (postdiscontinuation): 30 days

Long-term follow-up (postdiscontinuation): until death or study completion

**Reference Therapy, Dose, and Mode of Administration:** Erlotinib 150 mg administered orally as a tablet every 24 hours

### **Criteria for Evaluation:**

<u>Efficacy</u>: Efficacy assessments include imaging studies/tumor assessments, according to RECIST v. 1.1, performed every 8 weeks, and survival.

<u>Safety:</u> Safety will be evaluated based on recorded adverse events (AEs), physical examinations, vital sign measurements, and clinical laboratory assessments. Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA<sup>TM</sup>). Adverse events and clinical laboratory values will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.03 (NCI-CTCAE v. 4.03). <u>Health Outcomes:</u> Health outcomes will be assessed using standardized instruments, MDASI-LC and EQ-5D 5L. Investigators will report resource utilization such as concomitant medications, transfusions, radiation therapy, surgery, and treatment-related hospitalization days.

<u>Pharmacokinetics:</u> The plasma concentrations of LY2835219 and its metabolites LSN2839567, LSN3106726, and LSN3106729 will be measured for patients receiving LY2835219.

### <u>Biomarkers:</u>

*KRAS* mutation assessment: all tumor tissue samples (surgical resection, core needle biopsy, or fine needle aspirate) will be analyzed for *KRAS* mutation status by an investigational assay at the Study JPBK central laboratory. The same sample may also be used for evaluation of codons 12 and 13 via Sanger sequencing.

Other biomarkers: additionally, whole blood, plasma, and tissue samples will be tested for biomarkers relevant to LY2835219 and the disease state and to correlate these markers to clinical outcome and to LY2835219.

### **Statistical Methods:**

Statistical: The study will enroll approximately 550 patients in 3:2 randomization (330 patients in the LY2835219 arm and 220 patients in the erlotinib arm). The primary PFS analysis will be performed after 338 PFS events have occurred. In order to ensure an adequate number of patients have been enrolled for the analysis of OS, this analysis will not occur before 2 months after the study enrolls its last (approximately 550th) patient. The final OS analysis will occur when approximately 407 OS events have been observed. The study-wise alpha of .05 will be split between the endpoints: .005 for PFS and .045 for OS. A fallback procedure will be used. The test on PFS will occur first; if the test on PFS is significant, the alpha used for this test will be added to the .045 originally allocated to OS for a total of .05. This fallback procedure will maintain a study-wise alpha level of .05. While OS data are not anticipated to be mature at the time of the PFS analysis, .001 of the alpha allocated to OS will be spent at the time of the PFS analysis. Assuming a PFS hazard ratio (HR) of 0.67, this sample size yields approximately 80% statistical power to detect superiority of the LY2835219 arm over erlotinib arm with the use of a 2-sided log-rank test and a type I error of .005. If the true median PFS for the erlotinib arm is 2 months, then the HR of 0.67 amounts to an approximately 1-month improvement in median PFS for the LY2835219 arm under an additional assumption of exponential survival distribution. Assuming an OS HR of 0.75, this sample size yields approximately 80% statistical power to detect superiority of the LY2835219 arm over erlotinib arm with the use of a 2-sided log-rank test and a type I error of .045. If the true median OS for the erlotinib arm is 6.5 months, then the HR of 0.75 amounts to an approximately 2.2-month improvement in median OS for the LY2835219 arm under an additional assumption of exponential survival distribution.

Efficacy: Efficacy analyses will be based on the intention-to-treat (ITT) analysis set. This population is defined as all patients randomized to study treatment. For the co-primary endpoints of PFS and OS, the comparison of the survival curves between treatment groups will be conducted by a stratified log-rank test with the following stratification variables: number of prior chemotherapy regimens (1 versus 2), ECOG PS (0 versus 1), gender (male versus female), and *KRAS* mutation (GLY12CYS [G12C] vs. all others). In addition, the Kaplan-Meier method (Kaplan and Meier 1958) will be used to estimate the survival curves as well as survival rates at 3, 6, 9, and 12 months for each treatment group. As supportive analysis of OS and PFS, the Cox proportional hazard model will be used to estimate treatment HR and corresponding 95% confidence interval (CI) with Wald's test p-value after adjusting for the same randomization variables specified for the primary analysis. All randomized patients, according to the ITT principle, will be included in the analysis of this endpoint. An additional unstratified Cox regression model will be employed to explore the effects of prognostic variables, such as of the stratification variables and intrinsic/extrinsic factors, on treatment response.

<u>Safety:</u> All safety summaries and analyses will be based upon the Safety Population, defined as all enrolled patients receiving at least 1 dose of any study drug. Overall exposure to study drug, the numbers of patients completing each cycle, and the dose intensity will be summarized using descriptive statistics. An overall summary of AEs will be provided for AEs deemed by the investigator to be possibly related to study drug, and repeated for events regardless of study drug causality. Incidence rates of these events will be compared between treatment arms using Chi square test. CTCAE v 4.03 will be used to report AEs by CTCAE terms. Laboratory and nonlaboratory CTCAEs will be summarized by CTCAE term and maximum CTCAE grade, including the total for maximum Grade 3 and 4. The MedDRA Version 17.0 (or higher) will be used when reporting AEs by MedDRA terms. The MedDRA Lower Level Term will be used in the treatment-emergent computation. Treatment-emergent AEs will be summarized by System Organ Class (SOC) and by decreasing frequency of Preferred Term (PT) within SOC.

<u>Health Outcomes:</u> The MDASI-LC will be summarized for each assessment period. EQ-5D 5L responses for each item will be summarized by frequency and corresponding percentages. Descriptive statistics for the index and visual analog scale will be calculated.

<u>Pharmacokinetics:</u> Mean population PK parameters for LY2835219 in plasma (clearance, exposure, volume of distribution, and half-lives) and inter-individual PK variability will be computed using nonlinear mixed effect modeling (NONMEM). Covariate effects (such as age, weight, sex, creatinine clearance, and plasma protein levels) on the PK parameters of LY2835219 in plasma will also be investigated. The mean population PK properties of LY2835219 metabolites LSN2839567, LSN3106726, and LSN3106729 in plasma may also be analyzed by means of NONMEM.

### Biomarkers:

KRAS mutation assessment: Concordance (agreement) analysis will be performed on samples with valid KRAS status (mutation positive and mutation negative) using both the investigational assay and the reference method (Sanger sequencing). Measures of agreement between the investigational KRAS assay and the reference method, including positive percent agreement, negative percent agreement, and overall percent agreement, and their corresponding exact 2-sided 95% CI, will be estimated for the overall mutation status; that is, mutation detected or not detected for the 7 mutations of KRAS gene. A secondary agreement analysis between the investigational KRAS assay and the reference method will be performed for each of the tumor tissue sample types (surgical resection, fine needle aspirate, and core needle biopsy). The data will also be summarized for each of the 7 KRAS mutations separately.

Other biomarkers: the distributions of biomarkers will be summarized for the patient population for which samples are available. Associations between clinical endpoints and biomarker will be evaluated using data from patients who have an evaluable sample for each biomarker of interest, and such evaluation will be done on an individual marker basis.

# 3. Table of Contents

# A Randomized Phase 3 Study of LY2835219 plus Best Supportive Care versus Erlotinib plus Best Supportive Care in Patients with Stage IV NSCLC with a Detectable *KRAS* Mutation Who Have Progressed After Platinum-Based Chemotherapy

| Section | Page |
|---|---|
| 1. Protocol I3Y-MC-JPBK A Randomized Phase 3 Study of LY2835219 plus Best Supportive Care versus Erlotinib plus Best Supportive Care in Patients with Stage IV NSCLC with a Detectable <i>KRAS</i> Mutation Who Have Progressed After Platinum-Based Chemotherapy | 1 |
| 2. Synopsis | 2 |
| 3. Table of Contents | 6 |
| 4. Abbreviations and Definitions | 13 |
| 5. Introduction | 18 |
| 6. Objectives | 20 |
| 6.1. Primary Objective | 20 |
| 6.2. Secondary Objectives | 20 |
| 6.3. Exploratory Objectives | 20 |
| 7. Study Population | 21 |
| 7.1. Inclusion Criteria. | 21 |
| 7.2. Exclusion Criteria | |
| 7.2.1. Rationale for Exclusion of Certain Study Candidates | |
| 7.3. Discontinuations | |
| 7.3.1. Discontinuation of Patients | |
| 7.3.2. Discontinuation of Study Sites | |
| 8. Investigational Plan | |
| 8.1. Summary of Study Design | |
| 8.1.2. Extension Period | |
| 8.2. Discussion of Design and Control | |
| 9. Treatment. | |
| 9.1. Treatments Administered | |
| 9.2 Materials and Sunnlies | 30 |

| 9.3. Metho | od of Assignment to Treatment | 31 |
|---|---|---|
| 9.4. Select | ion and Timing of Doses | 31 |
| 9.4.1. | Special Treatment Considerations | 31 |
| 9.4.1.1. | Dose Adjustments and Delays | 31 |
| 9.4.1.1 | .1. LY2835219 | 31 |
| 9.4.1.1 | .2. Erlotinib | 32 |
| 9.5. Blindi | ng | 34 |
| 9.6. Conco | mitant Therapy | 34 |
| 9.6.1. I | Best Supportive Care | 35 |
| 9.6.1.1. | Palliative Radiotherapy | 35 |
| 9.6.1.2. | Antidiarrheal Agents | 35 |
| 9.6.1.3. | Antiemetic Agents | 36 |
| 9.6.1.4. | Analgesic Agents | 36 |
| 9.6.1.5. | Appetite Stimulants | 36 |
| 9.6.1.6. | Granulocyte-Colony Stimulating Factors (G-CSF) | 36 |
| 9.6.1.7. | Erythroid Growth Factors | 36 |
| 9.6.1.8. | Bone-Modifying Agents | 36 |
| 9.6.1.9. | Therapy for Febrile Neutropenia | 36 |
| 9.7. Treatr | nent Compliance | 37 |
| and the second s | Health Outcome/Quality of Life Measures, Safety | |
| Evaluation | ons, Sample Collection and Testing, and Appropriateness of | 20 |
| Evaluation Measures | ons, Sample Collection and Testing, and Appropriateness of ments | |
| Evaluation Measurer 10.1. Effica | ons, Sample Collection and Testing, and Appropriateness of ments | |
| Evaluation Measurer 10.1. Effica 10.1.1. | ons, Sample Collection and Testing, and Appropriateness of ments | 38 |
| Evaluation Measurer 10.1. Effica 10.1.1. I | ons, Sample Collection and Testing, and Appropriateness of ments cy Measures Efficacy Assessments at Baseline and during Study Treatment | 38 |
| Evaluation Measurer 10.1. Effica 10.1.1. In 10.1.2. In 10.1.2. | ons, Sample Collection and Testing, and Appropriateness of ments | 38 |
| Evaluation Measurer 10.1. Effica 10.1.1. If 10.1.2. If I | ons, Sample Collection and Testing, and Appropriateness of ments cy Measures Efficacy Assessments at Baseline and during Study Treatment Efficacy Assessments during the Study Period Postdiscontinuation Follow-Up | 38 38 |
| Evaluation Measurer 10.1. Effica 10.1.1. If 10.1.2. If 10.1.3. If 10.1.3. If 10.1.3. | ons, Sample Collection and Testing, and Appropriateness of ments cy Measures Efficacy Assessments at Baseline and during Study Treatment Efficacy Assessments during the Study Period Postdiscontinuation Follow-Up Primary Efficacy Measure | 38<br>38<br>39 |
| Evaluation Measurer 10.1. Effica 10.1.1. If 10.1.2. If 10.1.3. If 10.1.4. S | ons, Sample Collection and Testing, and Appropriateness of ments cy Measures Efficacy Assessments at Baseline and during Study Treatment Efficacy Assessments during the Study Period Postdiscontinuation Follow-Up Primary Efficacy Measure Secondary Efficacy Measures | 38<br>38<br>39<br>39 |
| Evaluation Measurer 10.1. Effica 10.1.1. If 10.1.2. If 10.1.3. If 10.1.4. State 10.2. Health | ons, Sample Collection and Testing, and Appropriateness of ments cy Measures Efficacy Assessments at Baseline and during Study Treatment Efficacy Assessments during the Study Period Postdiscontinuation Follow-Up Primary Efficacy Measure Secondary Efficacy Measures n Outcome/Quality of Life Measures | 38<br>38<br>39<br>39<br>40 |
| Evaluation Measurer 10.1. Effica 10.1.1. If 10.1.2. If 10.1.3. If 10.1.4. State 10.2. Health | ons, Sample Collection and Testing, and Appropriateness of ments cy Measures Efficacy Assessments at Baseline and during Study Treatment Efficacy Assessments during the Study Period Postdiscontinuation Follow-Up Primary Efficacy Measure Secondary Efficacy Measures n Outcome/Quality of Life Measures Patient-Reported Outcomes | |
| Evaluation Measurer 10.1. Effica 10.1.1. If 10.1.2. If 10.1.3. If 10.1.4. State 10.2. Health 10.2.1. If 10.2.1. If 10.2.1. | ons, Sample Collection and Testing, and Appropriateness of ments cy Measures Efficacy Assessments at Baseline and during Study Freatment Efficacy Assessments during the Study Period Postdiscontinuation Follow-Up Primary Efficacy Measure Secondary Efficacy Measures n Outcome/Quality of Life Measures Patient-Reported Outcomes MDASI-LC | 38<br>38<br>39<br>39<br>40<br>40<br>40 |
| Evaluation Measurer 10.1. Effica 10.1.1. If 10.1.2. If 10.1.3. If 10.1.4. State 10.2.1. If 10.2.1. If 10.2.1. If 10.2.1.1. If 10.2.1.2. | ons, Sample Collection and Testing, and Appropriateness of ments cy Measures Efficacy Assessments at Baseline and during Study Freatment Efficacy Assessments during the Study Period Postdiscontinuation Follow-Up Primary Efficacy Measure Secondary Efficacy Measures n Outcome/Quality of Life Measures Patient-Reported Outcomes MDASI-LC | 38<br>38<br>39<br>39<br>40<br>40<br>40 |
| Evaluation Measurer 10.1. Effica 10.1.1. If 10.1.2. If 10.1.3. If 10.1.4. State 10.2.1. If 10.2.1. If 10.2.1.1. If 10.2.1.2. If 10.2.1.2. If 10.2.2. If 10 | ons, Sample Collection and Testing, and Appropriateness of ments cy Measures Efficacy Assessments at Baseline and during Study Treatment Efficacy Assessments during the Study Period Postdiscontinuation Follow-Up Primary Efficacy Measure Secondary Efficacy Measures n Outcome/Quality of Life Measures Patient-Reported Outcomes MDASI-LC EQ-5D 5L | 38<br>38<br>39<br>39<br>40<br>40<br>40<br>40 |
| Evaluation Measurer 10.1. Effica 10.1.1. If 10.1.2. If 10.1.3. If 10.1.4. S 10.2. Health 10.2.1. If 10.2.1.1. 10.2.1.2. 10.2.2. If 10.3. Safety | ons, Sample Collection and Testing, and Appropriateness of ments cy Measures Efficacy Assessments at Baseline and during Study Treatment Efficacy Assessments during the Study Period Postdiscontinuation Follow-Up Primary Efficacy Measure Secondary Efficacy Measures n Outcome/Quality of Life Measures Patient-Reported Outcomes MDASI-LC EQ-5D 5L Resource Utilization | 38 38 38 39 40 40 40 40 41 |
| Evaluation Measurer 10.1. Effica 10.1.1. If 10.1.2. If 10.1.3. If 10.1.4. S 10.2. Health 10.2.1. If 10.2.1.1. 10.2.1.2. 10.2.2. If 10.3. Safety | ons, Sample Collection and Testing, and Appropriateness of ments cy Measures Efficacy Assessments at Baseline and during Study Treatment Efficacy Assessments during the Study Period Postdiscontinuation Follow-Up Primary Efficacy Measure Secondary Efficacy Measures a Outcome/Quality of Life Measures Patient-Reported Outcomes MDASI-LC EQ-5D 5L Resource Utilization Adverse Events | 38 38 38 39 40 40 40 40 41 41 42 |
| Evaluation Measurer 10.1. Effica 10.1.1. If 10.1.2. If 10.1.3. If 10.1.4. S 10.2. Health 10.2.1. If 10.2.1.2. 10.2.2. If 10.3. Safety 10.3.1. If 10.3.1. I | ons, Sample Collection and Testing, and Appropriateness of ments cy Measures Efficacy Assessments at Baseline and during Study Treatment Efficacy Assessments during the Study Period Postdiscontinuation Follow-Up Primary Efficacy Measure Secondary Efficacy Measures n Outcome/Quality of Life Measures Patient-Reported Outcomes MDASI-LC EQ-5D 5L Resource Utilization Pevaluations Adverse Events Serious Adverse Events | 38 38 38 39 40 40 40 41 41 41 42 |

| 10.3.2. | 1. Electrocardiograms | 45 |
|------------|---------------------------------------------------------|----|
| 10.3.3. | Safety Monitoring | 45 |
| 10.3.4. | Complaint Handling | 46 |
| 10.4. Sam | ple Collection and Testing | 46 |
| 10.4.1. | Samples for Study Qualification and Health Monitoring | 47 |
| 10.4.2. | Samples for KRAS Mutation Determination | 47 |
| 10.4.3. | Samples for Other Biomarkers | 48 |
| 10.4.3. | 1. Archived Tumor Tissue | 48 |
| 10.4.3. | 2. Blood Samples for Pharmacogenetic Evaluations | 48 |
| 10.4.3. | 3. Plasma Samples for Exploratory Biomarker Evaluations | 48 |
| 10.4.4. | Samples for Drug Concentration Measurements | |
| | Pharmacokinetics | |
| 10.5. App | propriateness of Measurements | 49 |
| 11. Data Q | uality Assurance | 50 |
| 11.1. Data | a Capture System | 50 |
| 12. Sample | Size and Statistical Methods | 51 |
| 12.1. Dete | ermination of Sample Size | 51 |
| 12.2. Stat | istical and Analytical Plans | 51 |
| 12.2.1. | General Considerations | 51 |
| 12.2.2. | Patient Disposition | 52 |
| 12.2.3. | Patient Characteristics | 52 |
| 12.2.4. | Concomitant Therapy | 52 |
| 12.2.4. | 1. Postdiscontinuation Therapy | 53 |
| 12.2.5. | Treatment Compliance | 53 |
| 12.2.6. | Primary Outcome and Methodology | 53 |
| 12.2.7. | Secondary Outcome and Methodology | 54 |
| 12.2.8. | Sensitivity Analysis | 55 |
| 12.2.9. | Pharmacokinetic Analyses. | 55 |
| 12.2.10. | Biomarker Analyses | 56 |
| 12.2.10 | 0.1. KRAS Mutation Assessment | 56 |
| 12.2.10 | 0.2. Other Biomarkers | 56 |
| 12.2.11. | Health Outcome/Quality of Life Analyses | 56 |
| 12.2.11 | I.1. MDASI-LC | 56 |
| | 1.2. Health State Utility | |
| 12.2.11 | 1.3. Use of Pain Medications | 57 |
| 12.2.12. | Safety Analyses | 57 |
| 12.2.13. | Subgroup Analyses | 58 |
| 12.2.14 | Interim Analyses | 58 |

| I3Y-MC-JPBK Clinical Protocol | Page 9 |
|---|---|
| 12.2.14.1. Safety Interim Analyses | 58 |
| 12.2.14.2. Efficacy Interim Analyses | 59 |
| 13. Informed Consent, Ethical Review, and Regulatory Considerations . | 60 |
| 13.1. Informed Consent. | 60 |
| 13.2. Ethical Review | 60 |
| 13.3. Regulatory Considerations | 61 |
| 13.3.1. Investigator Information | 61 |
| 13.3.2. Protocol Signatures | 61 |
| 13.3.3. Final Report Signature | 61 |
| 14. References | 62 |

# **List of Tables**

| Table | | Page |
|---|---|---|
| Table JPBK.9.1. | Treatment Regimens/Dosing Schedule | 30 |
| Table JPBK.9.2. | Dose Adjustments of LY2835219 for Study I3Y-MC-JPBK | 32 |
| Table JPBK.9.3. | Erlotinib Dose Reduction Schedule | 33 |
| Table JPBK.9.4. | Erlotinib Dose Modification Table. | 34 |
| Table JPBK.10.1. | Adverse Event and Serious Adverse Event Reporting Guidelines | 42 |
| Table JPBK.10.2. | Schedule for Electrocardiogram Collection | 45 |
| Table JPBK.12.1. | Alpha Allocation (2-Sided) for Progression-Free Survival and<br>Overall Survival | 53 |
| Table JPBK.12.2. | Rules for Determining Date of Progression or Censor for Progression-Free Survival. | 54 |
| Table JPBK.12.3. | World Health Organization Pain Scale | 57 |

# **List of Figures**

| Figure | | Page |
|------------------|-------------------------------------------|------|
| Figure JPBK.8.1. | Illustration of study design. | 26 |
| Figure JPBK.8.2. | Study period and extension period diagram | 28 |

# **List of Attachments**

| Attachment | | Page |
|---|---|---|
| Attachment 1. | Protocol JPBK Study Schedule | 64 |
| Attachment 2. | Protocol JPBK Clinical Laboratory Tests | 69 |
| Attachment 3. | Protocol JPBK Hepatic Monitoring Tests for Treatment-Emergent Abnormality | |
| Attachment 4. | Protocol JPBK ECOG Performance Status | 71 |
| Attachment 5. | Protocol JPBK RECIST Criteria 1.1 | 72 |
| Attachment 6. | Protocol JPBK Sampling Summary | 79 |
| Attachment 7. | Protocol JPBK Pharmacokinetic Sampling Schedule | 80 |
| Attachment 8. | Protocol JPBK Inducers and Strong Inhibitors of CYP3A4 or Substrates of CYP2B6 | 81 |

# 4. Abbreviations and Definitions

| Term | Definition |
|---|---|
| AE | adverse event |
| | Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. |
| ALT | alanine aminotransferase |
| ANC | absolute neutrophil count |
| ASCO | American Society of Clinical Oncology |
| assent | Agreement from a child or other individual who is not legally capable of providing consent, but who can understand the circumstances and risks involved in participating in a study (required by some institutional review boards [IRBs]). |
| AST | aspartate aminotransferase |
| audit | A systematic and independent examination of the trial-related activities and documents to determine whether the evaluated trial-related activities were conducted, and the data were recorded, analyzed, and accurately reported according to the protocol, applicable standard operating procedures (SOPs), good clinical practice (GCP), and the applicable regulatory requirement(s). |
| BOR | best overall response |
| BSC | best supportive care |
| CDK | p16INK4A-cyclin D-cyclin-dependent kinases |
| CI | confidence interval |
| CNS | central nervous system |
| collection database | A computer database where clinical trial data are entered and validated. |
| companion diagnostic | An in vitro diagnostic device (assay or test) that provides information that is essential for the safe and effective use of a corresponding therapeutic product |
| CRF/eCRF | case report form/electronic case report form |
| | Sometimes referred to as clinical report form: A printed or electronic form for recording study participants' data during a clinical study, as required by the protocol. |
| CRP | clinical research physician |
| | Individual responsible for the medical conduct of the study. Responsibilities of the CRP may be performed by a physician, clinical research scientist, global safety physician, or other medical officer. |

**CNS** central nervous system

**complaint** A complaint is any written, electronic, or oral communication that alleges deficiencies

related to the identity, quality, purity, durability, reliability, safety or effectiveness, or

performance of a drug or drug delivery system.

**compliance** Adherence to all the trial-related requirements, good clinical practice (GCP)

requirements, and the applicable regulatory requirements.

**CR** complete response

**CSR** clinical study report

**CT** computed tomography

CTCAE Common Terminology Criteria for Adverse Events

**CYP** cytochrome P450

**DCR** disease control rate

**DMC** data monitoring committee

**ECG** electrocardiogram

**ECOG** Eastern Cooperative Oncology Group

**EGFR** Epidermal growth factor receptor

end of trial End of trial is the date of the last visit or last scheduled procedure for the last patient.

enroll The act of assigning a patient to a treatment. Patients who are enrolled in the trial are

those who have been assigned to a treatment.

**enter** Patients entered into a trial are those who sign the informed consent form directly or

through their legally acceptable representatives.

**ERB** ethical review board

A board or committee (institutional, regional, or national) composed of medical and nonmedical members whose responsibility is to verify that the safety, welfare, and

human rights of the patients participating in a clinical trial are protected.

**EQ-5D 5L** European Quality of Life – 5 Dimensions – 5 Level

**extension period** The period between study completion and end of trial during which patients on study

therapy who continue to experience clinical benefit may continue to receive study

therapy until one of the criteria for discontinuation is met.

FDA US Food and Drug Administration

**FFPE** formalin-fixed paraffin-embedded

GLY12CYS: a mutation in codon 12 of the KRAS gene resulting in an amino acid

substitution from glycine to cysteine

**GCP** good clinical practice

**G-CSF** Granulocyte-Colony Stimulating Factors

**GPS** (Lilly) Global Patient Safety

**HIV** human immunodeficiency virus

**HR** hazard ratio

**IB** Investigator's Brochure

**ICF** informed consent form

**ICH** International Conference on Harmonisation

**Informed consent** A process by which a patient voluntarily confirms his or her willingness to participate

in a particular trial, after having been informed of all aspects of the trial that are relevant to the patient's decision to participate. Informed consent is documented by means of a

written, signed, and dated informed consent form.

interim analysis An interim analysis is an analysis of clinical trial data, separated into treatment groups,

that is conducted before the final reporting database is created/locked.

investigational

product

A pharmaceutical form of an active ingredient or placebo being tested or used as a

reference in a clinical trial.

**investigator** A person responsible for the conduct of the clinical trial at a trial site. If a trial is

conducted by a team of individuals at a trial site, the investigator is the responsible

leader of the team and may be called the principal investigator.

**ITT** intention-to-treat

The principle that asserts that the effect of a treatment policy can be best assessed by evaluating on the basis of the intention to treat a patient (that is, the planned treatment regimen) rather than the actual treatment given. It has the consequence that patients allocated to a treatment group should be followed up, assessed, and analyzed as members of that group irrespective of their compliance to the planned course of

treatment.

**KRAS** kirsten rat sarcoma

**legal representative** An individual, judicial, or other body authorized under applicable law to consent on

behalf of a prospective patient to the patient's participation in the clinical study.

Lilly Safety System Global safety database that tracks and reports serious adverse and spontaneous events

occurring while using a drug/drug delivery system.

**LLT** Lower Level Term

MD Anderson Symptom Inventory – Lung Cancer

Medical Dictionary for Regulatory Activities

MRI magnetic resonance imaging

NCI National Cancer Institute

**NONMEM** nonlinear mixed effect modeling

**NSCLC** non-small cell lung cancer

**OS** overall survival

**patient** A study participant who has the disease or condition for which the investigational

product is targeted.

**PD** progressive disease

**PET** positron emission tomography

**PK** pharmacokinetic

**PFS** progression-free survival

**PO** orally

**PR** partial response

**Pre-screen** The act of determining if an individual meets minimum requirements to be an

appropriate candidate for screening for a clinical study. In this study, prescreening involves diagnostic testing of an archived NSCLC tumor sample for mutations in codons 12 and 13 of the *KRAS* oncogene. Informed consent for this prescreening test shall be obtained; this consent may be separate from obtaining consent for the study.

**PS** performance status

PT Preferred Term

Q12H every 12 hours

QTc corrected QT interval

**RANKL** nuclear factor kappa B ligand

randomize the process of assigning patients to an experimental group on a random basis

**RECIST** Response Evaluation Criteria in Solid Tumors

**reporting database** A point-in-time copy of the collection database. The final reporting database is used to

produce the analyses and output reports for interim or final analyses of data.

**re-screen** to screen a patient who was previously declared a screen failure for the same study

**SAE** serious adverse event

**SAP** statistical analysis plan

**screen** The act of determining if an individual meets the requirements to become part of a pool

of potential candidates for participation in a clinical study. In this study, screening involves invasive or diagnostic procedures and/or tests (for example, x-rays, blood draws). Informed consent for these screening procedures and/or tests shall be obtained

screen failure patient who does not meet one or more criteria required for participation in a trial

**SD** stable disease

SmPC Summary of Product Characteristics

**SOC** System Organ Class

**study completion** This study will be considered complete after the final analysis of overall survival is

performed.

**SUSARs** suspected unexpected serious adverse reactions

**TEAE** treatment-emergent adverse event

Any untoward medical occurrence that either occurs or worsens at any time after treatment baseline and that does not necessarily have to have a causal relationship with

this treatment.

**TKI** tyrosine kinase inhibitor

**ULN** upper limits of normal

**US** United States

**VAS** visual analog scale

# A Randomized Phase 3 Study of LY2835219 plus Best Supportive Care versus Erlotinib plus Best Supportive Care in Patients with Stage IV NSCLC with a Detectable *KRAS*Mutation Who Have Progressed After Platinum-Based Chemotherapy

# 5. Introduction

Patients with metastatic non-small cell lung cancer (NSCLC) that harbor *KRAS* mutations (25%) have a poor prognosis compared to NSCLC patients who are *KRAS* wild-type (Guan et al. 2013). The p16INK4A-cyclin D-cyclin-dependent kinases (CDK) 4/6-retinoblastoma pathway is frequently dysregulated in NSCLC and therefore this pathway represents an attractive therapeutic target. Importantly, synthetic lethal interaction between *KRAS* mutation and CDK4 inhibition indicates a potential therapeutic application for CDK4/6 inhibitors in NSCLC (Puyol et al. 2010).

LY2835219 is a potent and selective small molecule inhibitor of CDK4/6. LY2835219 administered orally demonstrates single-agent activity in xenograft models of human NSCLC. In the Phase 1 study I3Y-MC-JPBA (JPBA), LY2835219 has shown acceptable safety/tolerability, as well as evidence of clinical activity in multiple tumor types. In addition, Study JPBA included a NSCLC expansion cohort that enrolled 57 patients with advanced and/or metastatic NSCLC. The *KRAS* status of the tumors from 53 of the 57 patients has been identified. For patients with *KRAS* mutant tumors (N=29), 16 patients had a Response Evaluation Criteria In Solid Tumors (RECIST) response of stable disease (SD) or better (disease control rate [DCR=55.2%]); for patient with *KRAS* wild-type tumors (N=24), 9 had a response of SD or better (DCR=37.5%).

In clinical trials, the most frequently reported adverse events (AEs) related to LY2835219 have been diarrhea, nausea, fatigue, and vomiting. These AEs have generally been low-grade events.

More information about the known and expected benefits, risks, and reasonably anticipated AEs of LY2835219 may be found in the Investigator's Brochure (IB). Information on AEs expected to be related to LY2835219 may be found in Section 7 (Development Core Safety Information) of the IB. Information on serious adverse events (SAEs) expected in the study population independent of drug exposure and that will be assessed by the sponsor in aggregate, periodically during the course of the study, may be found in Section 6 (Effects in Humans) of the IB.

More detailed information about the known and expected benefits and risks of erlotinib may be found in the following: Tarceva Package Insert or Summary of Product Characteristics (SmPC).

An investigational in vitro diagnostic medical device, or companion diagnostic, will be used to evaluate *KRAS* mutations in formalin-fixed paraffin-embedded (FFPE) NSCLC tumor tissue. The QIAGEN® *therascreen*® KRAS Rotor-Gene Q (RGQ) Polymerase Chain Reaction (PCR) Kit NSCLC is a real-time qualitative PCR assay used for the detection of 7 somatic mutations in codons 12 and 13 in the *KRAS* oncogene. Potential risks to patients have been evaluated by Eli

Lilly and Company's (Lilly's) Global Patient Safety (GPS). Physicians will consider each patient's disease, *KRAS* test result, and other factors to reach the appropriate therapeutic decision. No treatment decision shall be made solely on the basis of the *KRAS* test result. In the event LY2835219 would be administered to a patient for whom it is not indicated based on the result of the *KRAS* test result, there is no evidence from clinical studies indicating that this might cause or contribute to any serious harm of a patient, other than potentially delaying another treatment option for a patient. It is unlikely that an incorrect result would be generated by the in vitro diagnostic medical device and highly likely that an incorrect result would be detected by laboratory personnel.

Erlotinib is indicated for the treatment of patients with locally advanced or metastatic NSCLC after failure of at least 1 prior chemotherapy regimen (Tarceva United States [US] package insert [USPI], 2010). Unlike the use of erlotinib for first-line treatment of patients with NSCLC, second- and third-line treatment has no limitation with regard to epidermal growth factor receptor (EGFR) or KRAS mutation status. However, there has been some concern regarding the activity of erlotinib in treating NSCLC with KRAS mutations due to results from 3 studies. First, in the original BR-21 study, a subgroup evaluation of 30 patients with KRAS mutant tumors randomized between placebo and erlotinib demonstrated a nonsignificant better survival outcome in the placebo group (Zhu et al. 2008). Second, in TITAN, a second-line study of erlotinib versus chemotherapy, 35 patients with KRAS mutant tumors had inferior outcome on erlotinib compared to chemotherapy (Ciuleanu et al. 2012). Lastly, a meta-analysis of response rate showed numerically inferior response rate in patients with KRAS mutant tumors treated with EGFR tyrosine kinase inhibitors (TKIs, such as erlotinib and gefitinib) (Linardou et al. 2008). In the TAILOR study comparing docetaxel to erlotinib as second-line therapy, overall survival (OS) favored docetaxel treatment in patients with both KRAS wild-type and KRAS mutant tumors (hazard ratio [HR] = 0.79 and 0.81, respectively); similarly, progression-free survival (PFS) favored docetaxel (HR = 0.68 and 0.89) for KRAS wild-type and KRAS mutant, respectively (Garassino et al. 2013). There was not a significant treatment interaction based on KRAS status. However, the SATURN study of erlotinib maintenance therapy demonstrated that improved PFS was preserved in a subset of 90 patients with KRAS mutant tumors (HR = 0.77 erlotinib compared to placebo) (Brugger et al. 2011). Overall, the data remain conflicting and after extensive review of the literature, Langer stated, "KRAS mutation cannot be used at this time to preclude NSCLC patients from receiving anti-EGFR TKI's" (Langer 2011). The selection of treatment depends on the overall benefit/risk for the patient. Given the differences in toxicity profile for available treatments, and the limited treatment options for patients, erlotinib is an acceptable control arm as the only oral drug available for patients with lung cancer, and only approved drug for treatment of third-line patients.

The Phase 3 Study I3Y-MC-JPBK (JPBK) study will evaluate the clinical activity of LY2835219 plus best supportive care (BSC) versus erlotinib plus BSC for patients with Stage IV NSCLC whose tumors have a detectable *KRAS* mutation (specifically, in codons 12 or 13 of the *KRAS* oncogene as determined by an investigational assay at the Study JPBK central laboratory) and who have progressed after prior platinum based therapy and received 1 other prior therapy or are not eligible for further chemotherapy.

# 6. Objectives

# 6.1. Primary Objective

The co-primary objectives of this study are to compare LY2835219 plus BSC versus erlotinib plus BSC in patients with Stage IV NSCLC whose tumors have detectable *KRAS* mutations (specifically, in codons 12 or 13 of the *KRAS* oncogene as determined by an investigational assay at the Study JPBK central laboratory) and who have progressed after prior platinum-based therapy and 1 other prior therapy or are not eligible for further chemotherapy with respect to:

- progression-free survival (PFS)
- overall survival (OS)

# 6.2. Secondary Objectives

The secondary objectives of the study are to compare LY2835219 plus BSC to erlotinib plus BSC with respect to:

- overall response rate (complete response [CR] + partial response [PR])
- changes in patient-reported pain and disease-related symptoms collected via the MD Anderson Symptom Inventory (MDASI-LC) and changes in health status via European Quality of Life 5 Dimensions 5 Level (EQ-5D 5L).
- safety and tolerability
- resource utilization (for example, analgesic type, hospitalization, transfusion)
- the pharmacokinetic (PK)/pharmacodynamic properties of LY2835219

# 6.3. Exploratory Objectives

The exploratory objectives of the study are as follows:

• to explore biomarkers relevant to LY2835219 and the disease state and to correlate these markers to clinical outcome and to LY2835219

# 7. Study Population

Patients who do not meet the criteria for participation in this study (screen failure) may not be re-screened. Repeating laboratory tests (including re-test for *KRAS*) during the screening period does not constitute re-screening.

Prospective approval of protocol deviations to recruitment and enrollment criteria (also known as protocol waivers or exemptions) is not permitted.

### 7.1. Inclusion Criteria

Patients are eligible to be included in the study only if they meet all of the following criteria:

- [1] The patient must have confirmed diagnosis of stage IV NSCLC according to the American Joint Committee on Cancer Staging Handbook (Edge et al. 2009).
  - patients can have any T stage tumor, that is, any size primary with any amount of direct extension into surrounding structures,
  - any N stage tumor, that is, any LN spread in the chest, and
  - one or more of the following:
    - o cancer has spread to the opposite lung,
    - o cancer cell are found in a pleural effusion,
    - o cancer cells are found in a pericardial effusion, or
    - o cancer has spread to distant structures such as liver, bone, or brain.
- [2] availability of adequate FFPE tumor-derived material (tumor blocks or slides) from a biopsy, surgery or fine needle aspirate for analysis of *KRAS* mutation status. This sample should be the most recent available sample containing adequate material. Tumor sample requirements are described in Section 10.4.2. The sponsor will not request rebiopsy solely for the purpose of testing of *KRAS* status.
- [3] determined to have detectable mutations in codons 12 or 13 of the *KRAS* oncogene by an investigational assay at the Study JPBK central laboratory
- [4] The patient must have progressed after platinum-based chemotherapy (with or without maintenance therapy [see below]) AND have received 1 other prior chemotherapy for advanced and/or metastatic disease OR is judged by the physician as ineligible for further standard second-line chemotherapy.
  - Recurrent disease after adjuvant or neoadjuvant therapy, 1 additional prior regimen is allowed, so adjuvant or neoadjuvant therapy do not count as prior therapy for advance disease.
  - The patient may not have received prior EGFR-targeted therapy, including any multi-target TKIs, which may inhibit EGFR (for example, vandetanib) in any setting for NSCLC.
  - The patient may have received prior therapy with bevacizumab.
  - The patient may have received maintenance therapy. Maintenance treatment is defined as therapy given within 42 days after the last dose of platinum-based

- chemotherapy in patients that have not progressed (complete response, partial response, or stable disease) after platinum-based, first-line induction chemotherapy.
- [5] have measureable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1, Eisenhauer et al. 2009)
- [6] have a performance status (PS) of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) scale (see Attachment 3)
- [7] have discontinued all previous therapies for cancer (including chemotherapy, radiotherapy, immunotherapy, and investigational therapy) for at least 21 days for myelosuppressive agents or 14 days for nonmyelosuppressive agents prior to receiving study drug
- [8] recovered from the acute effects of therapy (treatment related toxicity resolved to baseline) except for residual alopecia
- [9] have adequate organ function, including:
  - hematologic: absolute neutrophil count (ANC) ≥1.5 × 10<sup>9</sup>/L, platelets ≥100 × 10<sup>9</sup>/L, and hemoglobin ≥8 g/dL. Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin until the day after the erythrocyte transfusion.
  - hepatic: bilirubin ≤1.5 × the upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤3.0 times ULN. For patients with hepatic metastases, ALT and AST equaling ≤5.0 times ULN are acceptable.
  - renal: serum creatinine within normal limits,  $\leq 1.5 \times ULN$
- [10] are  $\geq$ 18 years of age
- [11a] are a man and agree to use a reliable method of birth control and to not donate sperm during the study and for at least 3 months following the last dose of study drug(s) or country requirements, whichever is longer, OR
- [11b] are a woman of child-bearing potential who tests negative for pregnancy at the time of enrollment based on a serum pregnancy test and agrees to use a reliable method of birth control during the study and for 3 months following the last dose of the study drug(s) or country requirements, whichever is longer
- [12] have an estimated life expectancy of at least 12 weeks
- [13] have given written informed consent/assent prior to any study-specific procedures
- [14] are able to swallow oral medications
- [15] are reliable and are willing to follow study procedures

### 7.2. Exclusion Criteria

Patients will be excluded from the study if they meet any of the following criteria:

- [16] are currently enrolled in a clinical trial involving an investigational product or non-approved use of a drug or device (other than the study drug/device used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
- [17] have received treatment with a drug that has not received regulatory approval for any indication within 14 or 21 days of the initial dose of study drug for a nonmyelosuppressive or myelosuppressive agent, respectively
- [18] have previously completed or withdrawn from this study or any other study investigating LY2835219
- [19] have a personal history of any of the following conditions: presyncope or syncope of either unexplained or cardiovascular etiology, ventricular arrhythmia (including but not limited to ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest
- [20] have the presence of unstable central nervous system (CNS) metastasis. History of CNS metastasis or stable CNS metastases are allowed (no longer requiring active therapy such as steroid medications). Patients with a history of CNS metastases must have a brain scan (for example, MRI) within 28 days of randomization to document stability, even if there have been no changes in symptoms.
- [21] have a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission with no therapy for that disease for a minimum of 3 years
- [22] have serious preexisting medical conditions that, in the judgment of the investigator, would preclude participation in this study
- [23] females who are pregnant or lactating
- [24] have active bacterial, fungal, and/or known viral infection (for example, human immunodeficiency virus [HIV] antibodies, hepatitis B surface antigen, or hepatitis C antibodies). Screening is not required for enrollment.

# 7.2.1. Rationale for Exclusion of Certain Study Candidates

Exclusion Criterion [19] is necessary because the effects of LY2835219 on corrected QT (QTc) prolongation are unknown; these conditions may put the patient at additional risk. Exclusion Criterion [20] is necessary because patients with unstable CNS metastasis are not likely to receive sufficient study treatment, preventing a full assessment of the agents administered in this study. Exclusion Criterion [23] is necessary because the effects of LY2835219 on the developing fetus are unknown.

### 7.3. Discontinuations

### 7.3.1. Discontinuation of Patients

The criteria for enrollment must be followed explicitly. If the investigator site identifies a patient who did not meet enrollment criteria and who was inadvertently enrolled, the sponsor must be notified. If the sponsor identifies a patient who did not meet enrollment criteria and who was inadvertently enrolled, the investigator site will be notified. A discussion must occur between the sponsor clinical research physician (CRP) and the investigator to determine whether the patient may continue in the study, with or without study drug. Inadvertently enrolled patients may be maintained in the study and on study drug when the Lilly CRP agrees with the investigator that it is medically appropriate for that patient. The patient may not continue in the study with or without study drug if the Lilly CRP does not agree with the investigator's determination it is medically appropriate for the patient to continue. The investigator must obtain documented approval from the Lilly CRP to allow the inadvertently enrolled patient to continue in the study with or without study drug.

In addition, patients will be discontinued from the study drugs and/or from the study in the following circumstances:

- disease progression
- unacceptable toxicity
- the patient has had 2 dose reductions and experiences an AE that would cause a third dose reduction.
- the patient is significantly noncompliant with study procedures and/or treatment
- investigator decision
  - o the investigator decides that the patient should be discontinued from the study or study drug for any reason (for example, the patient becomes pregnant)
  - o if the patient, for any reason, requires treatment with another therapeutic agent that has been demonstrated to be effective for treatment of the study indication, discontinuation from the study drug occurs prior to introduction of the new agent
- patient decision
  - o the patient or the patient's designee (for example, parents or legal guardian) requests to be withdrawn from the study or study drug
- sponsor decision
  - Lilly stops the study or stops the patient's participation in the study for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and good clinical practice
- enrollment in any other clinical trial involving an investigational product or enrollment in any other type of medical research judged not to be scientifically or medically compatible with this study

The reason for and date of discontinuation will be collected for all patients. All randomized patients who discontinue regardless of whether or not they received study drug will have procedures performed as shown in the Study Schedule (Attachment 1).

# 7.3.2. Discontinuation of Study Sites

Study site participation may be discontinued if Lilly, the investigator, or the ethical review board (ERB) of the study site judges it necessary for medical, safety, regulatory, ethical, or other reasons consistent with applicable laws, regulations, and good clinical practice (GCP).

# 7.3.3. Discontinuation of the Study

The study will be discontinued if Lilly judges it necessary for medical, safety, regulatory, ethical, or other reasons consistent with applicable laws, regulations, and GCP.

# 8. Investigational Plan

# 8.1. Summary of Study Design

Study I3Y-MC-JPBK is a multicenter, randomized, open-label, parallel, comparator-controlled trial in patients with Stage IV NSCLC whose tumors have a detectable *KRAS* mutation in codons 12 or 13 by an investigational assay at the Study JPBK central laboratory and who have progressed after platinum-based chemotherapy and received 1 other prior therapy or are ineligible for further chemotherapy after platinum-based therapy.

Figure JPBK.8.1 illustrates the study design.



Abbreviations: ECOG = Eastern Cooperative Oncology Group; N = number of patients; NSCLC = non-small cell lung cancer; PD = progressive disease; PO = orally; PS = performance status; Q12H = every 12 hours; Q24H = every 24 hours.

### Figure JPBK.8.1. Illustration of study design.

Terms used to describe the periods during the study are defined below:

- **Pre-screening:** begins when the pre-screening informed consent form (ICF) is signed for evaluation of FFPE tissue and ends once the *KRAS* mutation status of the tissue is determined by the Study JPBK central laboratory (or at discontinuation, if the study ICF is not signed). Pre-screening for *KRAS* mutation status determination is optional. If pre-screening did not occur, determination of *KRAS* mutation status will occur at baseline.
- **Baseline:** begins when the study ICF is signed and ends at the first study treatment (or at discontinuation, if no treatment is given).
- **Study Period:** begins at the first study treatment and ends at study completion. The study period does not include the extension period.
  - o **Study Treatment Period:** begins at the first study treatment and ends when the patient and the investigator agree that the patient will no longer continue study

- treatment. The date of this agreement is to be reported on the case report form (CRF) as the Date of Discontinuation from study treatment.
- o **Postdiscontinuation Follow-Up:** begins the day after the patient and the investigator agree that the patient will no longer continue study treatment.

**Short-term follow-up** begins the day after the patient and the investigator agree that the patient will no longer continue study treatment and lasts approximately 30 days.

**Long-term follow-up** begins the day after short-term follow-up is completed and continues until the patient's death or overall study completion. During long-term follow-up, patients will have a follow-up visit every 60 days (±14 days).

- Extension Period: begins after study completion and ends at the end of trial. During the extension period, patients on study therapy who continue to experience clinical benefit may continue to receive study therapy until one of the criteria for discontinuation is met. The extension period includes extension period follow-up.
  - Extension period follow-up: begins 1 day after the patient and the investigator agree that the patient will no longer continue treatment in the extension period and lasts approximately 30 days.

# 8.1.1. Study Completion and End of Trial

This study will be considered complete (that is, the scientific evaluation will be complete [study completion]) following the final analysis of overall survival, as determined by Lilly. Investigators will continue to follow the study schedule for all patients until notified by Lilly that study completion has occurred.

"End of trial" refers to the date of the last visit or last scheduled procedure for the last patient (Figure JPBK.8.2). The end of trial occurs after study completion and after the last patient has discontinued study treatment and completed extension period follow-up (if applicable).



Abbreviations: OS = overall survival; PFS = progression-free survival.

a Lilly will notify sites when this begins and ends.

Figure JPBK.8.2. Study period and extension period diagram.

### 8.1.2. Extension Period

Patients receiving LY2835219 and experiencing ongoing clinical benefit may continue to receive LY2835219 in the extension period until 1 of the criteria for discontinuation is met (Section 7.3). Patients receiving erlotinib will be discontinued from the study and cross-over to LY2835219 is not allowed. Lilly will notify investigators when the extension period begins.

Patients who are in short-term follow-up when the extension period begins will continue in short-term follow-up until the 30-day short-term follow-up visit is completed. Long-term follow-up does not apply.

Patients who are in long-term follow-up when the extension period begins will be discontinued from long-term follow-up.

During the extension period, all AEs, SAEs, and study drug exposure will be reported on the CRF. Serious adverse events will also be reported to Lilly GPS (see Section 10.3.1). In the event that an SAE occurs, Lilly may request additional information (such as local laboratory results, concomitant medications, and hospitalizations) in order to evaluate the reported SAE.

Investigators will perform any other standard procedures and tests needed to treat and evaluate patients; however, the choice and timing of the tests will be at the investigator's discretion. Lilly will not routinely collect the results of these assessments.

# 8.2. Discussion of Design and Control

A randomized, controlled design is being used in this study. Randomization minimizes systematic bias in the selection and assignment of patients to study therapy and provides justification for inferential statistical methods to be used on data from this study. It is expected that LY2835219 will produce better efficacy outcomes than the control; therefore, a 3:2 randomization has been used in this study. Using an appropriate concurrent control arm enables direct statistical estimation of benefits and harms due to study therapy and minimizes bias in the assessment and interpretation of observed treatment effects. Patients will be stratified for differences in factors thought to be associated with clinical outcomes to further reduce the potential for bias and improve the power of the analyses.

### 9. Treatment

### 9.1. Treatments Administered

The following treatments will be administered in this study:

- Experimental Arm A: LY2835219 200 mg orally every 12 hours plus BSC on Days 1 to 28 of a 28-day cycle. The total daily dose of LY2835219 is 400 mg.
- Control Arm B: Erlotinib 150 mg orally every 24 hours plus BSC on Days 1 to 28 of a 28-day cycle.

Table JPBK.9.1 shows the treatment regimens.

Table JPBK.9.1. Treatment Regimens/Dosing Schedule

| Regimen | Period/Cycle | Dose Day 1-28 |
|-----------|------------------------|----------------|
| LY2835219 | Treatment/28-day cycle | 200 mg PO Q12H |
| Erlotinib | Treatment/28-day cycle | 150 mg PO Q24H |

Abbreviations: PO = orally; Q12H = every 12 hours; Q24H = every 24 hours.

The investigator or his/her designee is responsible for the following:

- explaining the correct use of the drugs and the planned duration of each individual's treatment to the patient, site personnel, and/or the patient's legal representative,
- verifying that instructions are followed properly,
- maintaining accurate records of study drug dispensing and collection,
- and returning all unused drug to Lilly or its designee at the end of the study.

**Note:** In some cases, sites may destroy the study drug if, during the investigator site selection, the evaluator has verified and documented that the site has appropriate facilities and written procedures to dispose clinical trial materials.

Patients will be instructed to contact the investigator as soon as possible if they have a complaint or problem with the study drug so that the situation can be assessed.

# 9.2. Materials and Supplies

LY2835219 will be supplied by Lilly as capsules for oral administration. LY2835219 capsules should be stored according to the temperature range listed on the product label, and should not be opened, crushed, or chewed.

Erlotinib will be supplied where required as tablets for oral consumption. Erlotinib should be stored according to the temperature range listed on the product label.

All study drug provided by Lilly will be labeled according to local country regulatory requirements. All medication should be kept out of the reach of children and stored in the original packaging/container provided.

# 9.3. Method of Assignment to Treatment

Patients who meet all criteria for enrollment will be randomly assigned to receive either LY2835219 or erlotinib at Visit 1.

Randomization will be stratified by the following factors:

- number of prior chemotherapy regimens (1 versus 2)
- performance status (0 versus 1)
- gender (male versus female)
- KRAS mutation (GLY12CYS [G12C] versus all others)

Assignment to treatment groups will be determined by a computer-generated random sequence using an interactive web response system.

The chosen stratification factors have been identified as variables with the foremost influence on the primary objective of OS. Randomization will be performed separately within each of the 16 strata (or cells) defined by all combinations of these 4 variables.

# 9.4. Selection and Timing of Doses

On Cycle 1 Day 1, only one 200-mg dose of LY2835219 will be taken. Chronic oral administration of LY2835219 will be initiated on Cycle 1 Day 2 and continue throughout every cycle. LY2835219 will be taken orally every 12 (±approximately 2) hours on Days 1 through 28 of a 28-day cycle, for a total of 56 doses per cycle. During all cycles, LY2835219 should be taken at approximately the same times each day. If a patient misses or vomits a dose, that dose should be omitted.

Erlotinib will be taken orally on Days 1 through 28 of a 28-day cycle, for a total of 28 doses per cycle. During all cycles, erlotinib should be taken at approximately the same time each day. If a patient misses or vomits a dose, that dose should be omitted.

A cycle is defined as the planned treatment interval of 28 days plus any subsequent delay prior to the start of the next cycle. A delay of a cycle due to holidays, weekends, bad weather, or other unforeseen circumstances will be permitted up to 7 days and not counted as a protocol deviation. No more than 28 days' worth of erlotinib or LY2835219 should be dispensed per cycle.

A patient may continue to receive study drug until he or she meets 1 or more of the specified reasons for discontinuation (as described in Section 7.3.1).

# 9.4.1. Special Treatment Considerations

# 9.4.1.1. Dose Adjustments and Delays

### 9.4.1.1.1. LY2835219

Before the start of each cycle, hematologic toxicity possibly related to LY2835219 must resolve to either baseline or at least Grade 2. If a patient experiences Grade 4 hematologic toxicity possibly related to LY2835219, then dosing must be suspended (until the toxicity resolves to

either baseline or at least Grade 2) and the dose of LY2835219 must be reduced as outlined in Table JPBK.9.4.

Before the start of each cycle, nonhematologic toxicity (except alopecia and fatigue) possibly related to LY2835219 must resolve to either baseline or at least Grade 1. Refer to Section 9.6.1.2 for guidance and supportive measures of diarrhea toxicity possibly related to LY2835219. If a patient experiences  $\geq$ Grade 3 nonhematologic toxicity possibly related to LY2835219, then dosing must be suspended (until the toxicity resolves to either baseline or at least Grade 1) and the dose of LY2835219 must be reduced as outlined in Table JPBK.9.2.

If a patient experiences persistent or recurrent Grade 2 nonhematologic toxicity (such as diarrhea, as outlined in Section 9.6.1.2) possibly related to LY2835219 that does not resolve with maximal supportive measures within 7 days to either baseline or Grade 1, then dosing may be suspended (until the toxicity resolves to either baseline or at least Grade 1) and the dose of LY2835219 may be reduced as outlined in Table JPBK.9.2.

The start of a cycle may be delayed to allow sufficient time for recovery from toxicity possibly related to study drug. Patients not recovering from such toxicity within 14 days beyond the last day of the prior cycle will be considered for discontinuation from the study.

If a patient receiving the 100-mg dose of LY2835219 requires a further dose reduction, the patient should be discontinued from study treatment. If a patient who, in the judgment of the investigator, is receiving clinical benefit from study therapy requires further dose reduction than is outlined in Table JPBK.9.2, then the investigator must discuss with the Lilly CRP prior to any further dose reduction.

Dose omissions are allowed within a cycle. If a patient requires omission of more than 25% of doses during a cycle for tolerability, then treatment may continue if the investigator determines the patient is receiving clinical benefit. If the patient does well after a dose reduction and is receiving clinical benefit, the investigator may contact the Lilly CRP to discuss possible dose re-escalation. After re-escalation, subsequent dose adjustments should be based on the dose of LY2835219 that the patient is currently receiving.

Table JPBK.9.2. Dose Adjustments of LY2835219 for Study I3Y-MC-JPBK

| Dose Adjustment | Oral Dose | Frequency |
|-----------------|-----------|----------------|
| 0 | 200 mg | Every 12 hours |
| 1 | 150 mg | Every 12 hours |
| 2 | 100 mg | Every 12 hours |

### 9.4.1.1.2. Erlotinib

Patients should be treated following the recommendations, warnings, and precautions given for erlotinib in the SmPC of erlotinib. Patients receiving erlotinib can have the erlotinib dose reduced if the toxicity is specifically attributable to erlotinib.

The daily dose of erlotinib will be decreased in 50-mg decrements to a minimum dose of 50 mg daily (Table JPBK.9.3). Re-escalation of erlotinib dosing is allowed at the investigator's

discretion, except after Grade 3 diarrhea when re-escalation is not allowed. Dose reductions must be documented within the current cycle so that treatment compliance can be determined.

In addition to the common erlotinib toxicities in Table JPBK.9.4, if a patient experiences other Grade 3 or 4 events that are considered at least possibly related to erlotinib, erlotinib administration may be omitted until the event resolves. If dosing with erlotinib is delayed for more than 14 consecutive days, patient dosing with erlotinib should be discontinued.

- If the event resolves to ≤ Grade 1 or baseline, the patient may restart erlotinib treatment at a reduced dose (Table JPBK.9.3).
- If the event has not resolved to ≤ Grade 1 or baseline within 7 days, or another AE occurs during therapy at the reduced dose, a second dose reduction is permitted at the investigator's discretion.

If the patient does not tolerate at least the 50-mg daily erlotinib dose, erlotinib must be discontinued.

Table JPBK.9.3. Erlotinib Dose Reduction Schedule

| Dose Adjustment | Oral Dose | Frequency |
|-----------------|------------|-----------|
| 0 | 150 mg/day | Daily |
| 1 | 100 mg/day | Daily |
| 2 | 50 mg/day | Daily |

Table JPBK.9.4 shows the dose modification criteria and guidelines for management of common erlotinib toxicities.

Table JPBK.9.4. Erlotinib Dose Modification Table

| Event and Gradea | <b>Erlotinib Dose Modifications</b> | <b>Guidelines for Management</b> |
|---|---|---|
| Pulmonary Events | | |
| All grades (acute onset of new or progressive pulmonary symptoms such as dyspnea, cough, or fever) | Interrupt, pending the diagnostic<br>evaluation; if interstitial lung disease is<br>diagnosed, discontinue study treatment | |
| | and institute appropriate treatment | |
| Diarrhea | | |
| Grade 1 | None | Consider loperamide: 4 mg at first onset, followed by 2 mg every 2 to 4 hours until diarrheafree for 12 hours |
| Grade 2 | Reduce if diarrhea persists over 48 to 72 hours despite optimal medical management | Manage as for Grade 1 |
| Grade 3 or any grade unresponsive to loperamide, or diarrhea that causes dehydration | Interrupt until resolution to Grade ≤1 and restart at next reduced dose; do not re-escalate | Manage as for Grade 1 |
| Grade 4 | Discontinue erlotinib treatment | Manage as for Grade 1 |
| Rash | | - |
| Tolerable rash (Grade 2 or 3) | None | Any of the following:<br>minocycline, topical tetracycline,<br>topical clindamycin, topical silver<br>sulfadiazine, diphenhydramine,<br>oral prednisone (short course) |
| Intolerable rash | Consider interruption or dose reduction if unresponsive to symptomatic management. | Manage as for Grade 1 |
| Grade 4 | Discontinue erlotinib treatment | Manage as for Grade 1 |

Abbreviations: CTCAE = Common Terminology Criteria for Adverse Events; NCI = National Cancer Institute. a CTCAE (Version 4.03; NCI 2009).

# 9.5. Blinding

This is an open-label study.

# 9.6. Concomitant Therapy

Appropriate documentation of all forms of premedications, supportive care, concomitant medications, and supplements must be captured at each visit in the CRF. Concomitant medications and supportive care therapies must also be documented at the time of discontinuation and at the 30-day short-term follow-up visit.

The results from an in vitro human recombinant cytochrome P450 (CYP) phenotyping study indicate that oxidative metabolism of LY2835219 is primarily catalyzed by CYP3A4. However, the extent of oxidative metabolism responsible for the systemic clearance of LY2835219 in

humans is presently unknown. Based on these in vitro findings, grapefruit juice as well as inducers (for example, phenytoin or carbamazepine) and strong inhibitors of CYP3A4 should be substituted or avoided if possible (Attachment 8). In addition, in vitro studies in primary cultures of human hepatocytes indicate that LY2835219 might inhibit the metabolism of CYP2B6 substrate drugs in vivo in human. Based on this finding, sensitive CYP2B6 substrates such as bupropion and efavirenz should be substituted or avoided if possible (Attachment 8).

Erlotinib is also metabolized predominantly by CYP3A4; therefore, grapefruit juice as well as inducers (for example, phenytoin or carbamazepine) and strong inhibitors of CYP3A4 should be substituted or avoided if possible (Attachment 8).

# 9.6.1. Best Supportive Care

Palliative and supportive care for other disease-related symptoms and for toxicity associated with treatment will be offered to all patients on this trial. Supportive care measures may include but are not limited to antidiarrheal agents, antiemetic agents, opiate and nonopiate analgesic agents, appetite stimulants, and granulocyte and erythroid growth factors. Details of interventions (for example, medications such as sedatives, antibiotics, analgesics, antihistamines, steroids, or erythroid-stimulating agents), procedures (for example, paracentesis or thoracentesis), or blood products (for example, blood cells, platelets, or fresh frozen plasma transfusions) should be recorded on the electronic case report forms (eCRFs). If it is unclear whether a therapy should be regarded as supportive care, the investigator should consult the Lilly CRP. Use of any supportive care therapy should be reported on the CRFs. Guidelines regarding the use of other specific supportive care agents are presented below.

Additional concurrent chemotherapy, radiation therapy (except as noted in Section 9.6.1.1), biologic response modifiers, or other investigational agents may not be administered to patients on this study.

### 9.6.1.1. Palliative Radiotherapy

Palliative radiotherapy, unless required due to progressive disease, is permitted during the study.

### 9.6.1.2. Antidiarrheal Agents

Diarrhea may influence tolerability of LY2835219. During therapy with LY2835219, early treatment with antidiarrheal agents (for example, loperamide) is recommended immediately after the first loose stool and should be continued until loose bowel movements cease for 12 hours.

For patients who experience Grade 2 diarrhea lasting more than 48 hours despite maximal treatment with antidiarrheal agents or for patients who experience ≥Grade 3 diarrhea, withhold LY2835219 until diarrhea resolves to Grade 1 or less, and then resume LY2835219 with appropriate dose reduction according to Table JPBK.9.2.

In the event of Grade 3 or 4 diarrhea, supportive measures may include hydration, loperamide, octreotide, and other antidiarrheals. If diarrhea is severe (that is, requires intravenous hydration) and/or associated with fever or severe (Grade 3 or 4) neutropenia, broad-spectrum antibiotics must be prescribed. Patients with Grade  $\geq$ 3 diarrhea or any diarrhea associated with Grade  $\geq$ 3 nausea or vomiting should be considered for hospitalization for intravenous hydration and
correction of electrolyte imbalance. Events that require a patient to be hospitalized are considered SAEs (see Section 10.3.1.1).

Guidance for the management of diarrhea in patients receiving erlotinib is given in Table JPBK.9.4.

#### 9.6.1.3. Antiemetic Agents

The use of antiemetic agents is permitted during this study and at the discretion of the investigator. However, it is recommended to follow the guidelines of the Multinational Association of Supportive Care in Cancer and American Society of Clinical Oncology (ASCO); dexamethasone may be sufficient, but 5-HT3 antagonists and NK1 antagonists may be used (Kris et al. 2006; Gralla et al. 2010).

#### 9.6.1.4. Analgesic Agents

The use of analgesic agents (other than non-steroidal anti-inflammatory drugs) is permitted at the discretion of the investigator.

#### 9.6.1.5. Appetite Stimulants

The use of appetite stimulants is permitted at the discretion of the investigator. Acceptable agents include, but are not limited to, megestrol acetate and dronabinol.

#### 9.6.1.6. Granulocyte-Colony Stimulating Factors (G-CSF)

The use of granulocyte-colony stimulating factor (G-CSF) is permitted during investigational therapy at the discretion of the investigator. G-CSF or similar agents are strongly recommended following Grade 3 or 4 neutropenia of duration >5 days or following any incidence of febrile neutropenia (ANC <1.0 x  $10^3/\mu$ L [1.0 x  $10^9$ /L] with a single temperature  $\ge 38.3^\circ$ C or a sustained temperature of  $\ge 38.0^\circ$ C for >1 hour).

#### 9.6.1.7. Erythroid Growth Factors

The use of erythroid-stimulating factors (for example, erythropoietin) is permitted at the discretion of the investigator based on ASCO and FDA guidelines (Rizzo et al. 2008; FDA 2009).

#### 9.6.1.8. Bone-Modifying Agents

The use of approved bone-modifying agents (for example, bisphosphonates or receptor activator of nuclear factor kappa B ligand [RANKL] targeting agents) is allowed on study if a patient had initiated treatment with such agents at least 14 days prior to randomization. Patients who started the study while receiving bisphosphonates or RANKL targeted agents are not allowed to switch treatments (for example, replace bisphosphonates with denosumab) during study treatment. Patients are not permitted to begin treatment with bisphosphonates or RANKL-targeted agents while receiving study treatment.

#### 9.6.1.9. Therapy for Febrile Neutropenia

Patients experiencing febrile neutropenia, especially with diarrhea or dyspnea, should be managed in a hospital setting according to standard procedures, with the urgent initiation of intravenous antibiotic therapy. Events that require a patient to be hospitalized are considered SAEs (see Section 10.3.1.1).

#### 9.7. Treatment Compliance

Patient compliance with study drug will be assessed at each visit. Compliance will be assessed by counting returned tablets/capsules. Patients may use a diary to record study drug intake.

Patients who are significantly noncompliant will be discontinued from the study. Unless required secondary to toxicity, a patient will be considered significantly noncompliant if he or she misses 7 or more consecutive days of study drug (full doses), or more than 25% of the cumulative days of study drug (full doses) during a cycle. Persistent noncompliance may be a reason for discontinuation from study therapy. Similarly, a patient will be considered significantly noncompliant if he or she is judged by the investigator to have intentionally or repeatedly taken more than the prescribed amount of medication.

# 10. Efficacy, Health Outcome/Quality of Life Measures, Safety Evaluations, Sample Collection and Testing, and Appropriateness of Measurements

Written informed consent must be obtained prior to any study-specific pretreatment evaluations.

Study procedures related to efficacy, safety, health outcome/quality of life measures, sample collection, and testing assessments and their timing are described in the sections below and shown in the Study Schedule (Attachment 1).

## 10.1. Efficacy Measures

## 10.1.1. Efficacy Assessments at Baseline and during Study Treatment

Within 28 days before randomization, baseline tumor measurements will be performed on each patient. Computed tomography (CT), including spiral CT, scans, and magnetic resonance imaging (MRI) are the preferred methods of measurement. Tumor assessments should include the chest and abdominal region.

The CT portion of a positron emission tomography (PET)-CT scan may be used as a method of response assessment if the site can document that the CT is of identical diagnostic quality to a diagnostic CT (with intravenous and oral contrast). A PET scan alone or as part of a PET-CT may be performed for additional analyses but cannot be used to assess response according to RECIST.

The method of assessment used at baseline must be used consistently for tumor assessment and must be repeated every other cycle, beginning with Cycle 3 Day 1. If a cycle is delayed, tumor assessment should be concurrent with Day 1 of the new cycle.

Responses (CR or PR) must be confirmed no less than 28 days from the first evidence of response. Thereafter, a responding patient should be followed every other cycle until objective progression is observed.

For patients continuing treatment after study completion (that is, during the extension phase), efficacy assessments (frequency and type of assessments) will be at the discretion of the investigator, based on the standard of care.

## 10.1.2. Efficacy Assessments during the Study Period Postdiscontinuation Follow-Up

Postdiscontinuation follow-up during the study period will be conducted as described in the Study Schedule (Attachment 1).

For those patients who discontinue study treatment without objectively measured progressive disease (PD), the investigative sites will continue to monitor patients and periodically evaluate tumor response every 8 weeks by the same method used at baseline until the patient has objective disease progression, or study completion. After the patient has objective disease progression,

radiologic tests are no longer required and the patient will be followed up approximately every 60 days ( $\pm 14$  days) until the patient's death or overall study completion.

Response (CR or PR) should be confirmed before the initiation of additional anticancer therapy. However, initiation of new therapy should not be delayed solely to confirm response.

Efficacy assessments (frequency and type of assessments) for patients still on treatment during the extension phase will be at the discretion of the investigator, based on the standard of care.

## 10.1.3. Primary Efficacy Measure

This study has co-primary efficacy measures of PFS and OS.

Progression-free survival will be defined as the time from randomization until the first evidence of objective progression as defined by RECIST v1.1 (Eisenhauer et al. 2009), or death from any cause, whichever is earlier. Patients who are not known to have either progressed or died at the time of analysis will be censored at the day of their last radiographic tumor assessment, if available, or the date of randomization if no postbaseline radiographic assessment is available. The detailed censoring rules are described in Table JPBK.12.2.

The primary PFS analysis will be based on the local investigator's tumor assessments.

Lilly or its designee will collect and store all tumor measurement images on all enrolled patients throughout the study. A central review of imaging scans may be performed by Lilly or its designee.

Overall survival duration is measured from the date of randomization to the date of death from any cause. For each patient who is not known to have died as of the data-inclusion cutoff date for a particular analysis, OS will be censored for that analysis at the date of last contact prior to the data inclusion cutoff date (contacts considered in the determination of last contact date include adverse event date, lesion assessment date, visit date, and last known alive date).

## 10.1.4. Secondary Efficacy Measures

The secondary efficacy measure is response as defined by RECIST v1.1 (Eisenhauer et al. 2009) provided in Attachment 5. A responder is defined as any patient who exhibits a confirmed CR or PR.

Best response is determined from the sequence of responses assessed.

A second assessment must be performed ≥28 days after the first evidence of response. The next scheduled scan at 56 days (8 weeks) would qualify for response confirmation. Two objective status determinations of CR before progression are required for a best response of CR. Two determinations of PR or better before progression, but not qualifying for a CR, are required for a best response of PR. Best response of SD is defined as disease that does not meet the criteria for CR, PR, or PD and has been evaluated at least 1 time, at least 6 weeks after the start of study treatment.

Best response will be derived to encompass all tumor assessments from baseline until the earliest of objective progression or start of new anticancer therapy. Any responses observed after objective progression or the start of new anticancer therapy are excluded from the determination of best response.

The date of first documented objective disease progression must be recorded on the CRF even if it occurs after the patient has started a new therapy.

### 10.2. Health Outcome/Quality of Life Measures

## 10.2.1. Patient-Reported Outcomes

Patient-reported outcomes will be measured using standardized instruments, MDASI-LC and EQ-5D 5L.

Patient-reported questionnaires should be completed by patients when a language translation is available in which the patient is fluent or literate.

At each time point identified in the Schedule of Events (Attachment 1), a paper copy of the questionnaire should be administered to the patient prior to extensive interaction with site staff and study drug administration.

#### 10.2.1.1. MDASI-LC

The MDASI-LC (Mendoza et al. 2011) is a 22-item instrument that includes 13 core symptoms, 6 core interference items, and 3 lung-specific symptoms (coughing, constipation, and sore throat). An additional MDASI page will include 11 exploratory items that are not a standard part of the MDASI-LC instrument. Advanced lung cancer is a leading source of brain metastases, and symptoms related to brain metastases are described by 8 of these exploratory items (weakness on 1 side of body, difficulty understanding, difficulty speaking, seizures, difficulty concentrating, vision, change in appearance, and irritability). These 8 exploratory items for this study are also included as brain-specific items in the MDASI-Brain Tumor instrument. The remaining 3 exploratory items address an additional brain symptom (headache) and expected treatment-related toxicities (diarrhea, rash, or skin change).

"Worst pain" is the first MDASI-LC item, and use of pain medication will be assessed in conjunction with the MDASI-LC assessment as described in Section 10.2.2.

Responses for the MDASI-LC items are captured through the use of 11-point numeric rating scales anchored at 0 (*not present* or *does not interfere*) and ranged through 10 (*as bad as you can imagine* or *completely interferes*). The MDASI-LC recall period is 24 hours, and typical completion time for this instrument is less than 5 minutes.

#### 10.2.1.2. EQ-5D 5L

The EuroQol 5-Dimension 5 Level (EQ-5D 5L) is a self-reported standardized measure of health status, and will allow for comparison with other tumor types and disease states (Janssen et al. 2008).

Specifically, this questionnaire is included in this trial to evaluate health-state utilities associated with advanced lung cancer. These utility measures are an important input for economic evaluations concerning the value of treatment interventions.

The EQ-5D 5L is designed to be used in conjunction with other patient-reported measures. Patients will complete the 5-dimension (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), 5-level (no problem, slight, moderate, severe, or extreme problem) assessment according to the Study Schedule (Attachment 1). A visual analog scale "thermometer" measures current health state. EQ-5D 5L responses may be incorporated into cost utility analyses and will be summarized in the clinical study report (CSR).

Administration is preferably scheduled after the MDASI-LC, and before extensive contact with study personnel or clinicians, which could result in biased patient response. The recall period is "today." The EQ-5D 5L is designed for self-completion by respondents and expected completion time is 1 to 2 minutes.

#### 10.2.2. Resource Utilization

Investigators will be asked to report the use of **all** concomitant medications (in particular, analgesics, bisphosphonates, and RANK-L targeted agents), blood product transfusions, radiation therapy, surgery, and hospitalization days.

Data on each individual prescription and over-the-counter analgesic medication will be recorded on the Concomitant Medication eCRF. The use of pain medications from the previous visit should be reviewed with the patient at each subsequent visit. Any changes to analgesic use based on this information should be recorded on the Concomitant Medication eCRF, and the term "any changes" includes new or stopped analgesics. Data on neurosurgical blocks will be recorded on the analgesic and/or surgery forms as appropriate. This information should be collected during the study and at the 30-day follow-up visit.

## 10.3. Safety Evaluations

Investigators are responsible for monitoring the safety of patients who have entered this study and for alerting Lilly or its designee to any event that seems unusual, even if this event may be considered an unanticipated benefit to the patient.

Investigators must document their review of each laboratory safety report.

The investigator is responsible for the appropriate medical care of patients during the study.

The investigator remains responsible for following, through an appropriate health care option, AEs that are serious, considered related to the study, or that caused the patient to discontinue before completing the study. The patient should be followed until the event is resolved or explained. Frequency of follow-up evaluation is left to the discretion of the investigator.

The timing of all safety evaluations is shown in the Study Schedule (Attachment 1). Table JPBK.10.1 presents a summary of AE and SAE reporting guidelines. Table JPBK.10.1 also shows which database or system is used to store AE and SAE data.

Х

X

x

X

**Lilly Safety** Collection Period Types of AEs/SAEs to be Reported **Database System** Baseline (pretreatment) Preexisting conditions X All AEs X SAEs related to protocol procedures X Study treatment period All AEs X All SAEs X Х 30-day short-term All AEs X postdiscontinuation follow-up All SAEs Х Long-term postdiscontinuation All SAEs related to protocol procedures follow-up or study drug Extension period All AEs X

All SAEs related to protocol procedures

or study drug that the investigator

Table JPBK.10.1. Adverse Event and Serious Adverse Event Reporting Guidelines

Abbreviations: AEs = adverse events; SAEs = serious adverse events.

All SAEs

All AEs

All SAEs

becomes aware of

#### 10.3.1. Adverse Events

participating in the study (that is, no

longer receiving study therapy and

Extension period follow-up

After the patient is no longer

no longer in follow-up)

Lilly has standards for reporting AEs that are to be followed regardless of applicable regulatory requirements that may be less stringent. A clinical study AE is any untoward medical event associated with the use of a drug in humans, whether or not it is considered related to that drug.

Lack of drug effect is not an AE in clinical trials, because the purpose of the clinical trial is to establish drug effect.

Any clinically significant findings from electrocardiograms (ECGs; for example, QTc prolongation), labs, vital sign measurements, other procedures, and so on that result in a diagnosis should be reported to Lilly or its designee. All non-clinically significant findings must be documented in the patient record as not clinically significant and therefore will not be documented in the eCRF.

Cases of pregnancy that occur during maternal or paternal exposures to study drug should be reported. Data on fetal outcome and breast-feeding are collected for regulatory reporting and drug safety evaluation.

Study site personnel will record the occurrence and nature of each patient's preexisting conditions, including clinically significant signs and symptoms of the disease under treatment in the study. All non-clinically significant findings must be documented in the patient record as not clinically significant and therefore will not be documented in the eCRF.

After the study ICF is signed, site personnel will record the occurrence and nature of any AEs and any change in the preexisting condition(s). All AEs related to protocol procedures are reported to Lilly or its designee.

In addition, all AEs occurring after the patient receives the first dose of study drug must be reported to Lilly or its designee via eCRF.

Investigators will be instructed to report to Lilly or its designee their assessment of the potential relatedness of each AE to protocol procedure or study drug via eCRF.

The investigator will decide whether he or she interprets the observed AEs as related to disease, to the study drug, study procedure, or other concomitant treatment or pathologies. To assess the relationship of the AE to the study drug or procedure, the following terminologies are defined:

- **Probably related**: a direct cause and effect relationship between the study treatment and the AE is likely
- **Possibly related**: a cause and effect relationship between the study treatment and the AE has not been demonstrated at this time and is not probable, but is also not impossible
- **Does not know:** the investigator cannot determine
- **Not related**: without question, the AE is definitely not associated with the study treatment

The investigator should classify all "probably related," "possibly related," or "does not know" AEs and SAEs as related to study drug/study procedure.

Patients will be evaluated for AEs at each visit and will be instructed to call their physician to report any AEs between visits.

The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03 will serve as the reference document for choosing appropriate terminology for, and grading the severity of, all AEs and other symptoms. For AEs without matching terminology within the NCI-CTCAE v 4.03 criteria, the investigator will be responsible for selecting the appropriate system organ class and assessing severity grade based on the intensity of the event.

In addition to collecting the AE verbatim and the CTCAE severity grade, AE verbatim text will also be mapped by Lilly or its designee to corresponding terminology within the Medical Dictionary for Regulatory Activities (MedDRA) dictionary.

If a patient's dosage is reduced or treatment is discontinued as a result of an AE, study site personnel must clearly report to Lilly or its designee via eCRF the circumstances and data leading to any such dosage reduction or discontinuation of treatment.

#### 10.3.1.1. Serious Adverse Events

An SAE is any adverse event from this study that results in one of the following outcomes:

- death
- a life-threatening experience (that is, immediate risk of dying)

- persistent or significant disability/incapacity
- initial or prolonged inpatient hospitalization
- congenital anomaly/birth defect
- considered significant by the investigator for any other reason

Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious adverse drug events when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

Serious adverse event collection begins after the patient has signed the study ICF and has received study drug. If a patient experiences an SAE after signing informed consent, but prior to receiving study drug, the event will not be reported as serious unless the investigator feels the event may have been caused by a protocol procedure.

Data on SAEs that occur before the end of trial will be stored in the collection database and the Lilly Safety System.

Study site personnel must alert Lilly or its designee of any **serious** adverse event (SAE) within 24 hours of investigator awareness of the event via a sponsor-approved method. If alerts are issued via telephone, they are to be immediately followed with official notification on study-specific SAE forms.

This 24-hour notification requirement refers to the initial SAE information and all follow-up SAE information.

Planned surgeries should not be reported as SAEs unless the underlying medical condition has worsened during the course of the study.

Planned hospitalizations or procedures for preexisting conditions that are already recorded in the patient's medical history at the time of study enrollment should not be considered SAEs. Hospitalization or prolongation of hospitalization without a precipitating clinical AE (for example, for the administration of study therapy or other protocol-required procedure) should not be considered SAEs

Serious adverse events due to disease progression, including death, should not be reported unless the investigator deems them to be possibly related to the study drug.

If an investigator becomes aware of an SAE occurring after the patient's participation in the trial has ended, and the investigator believes that the SAE is related to a protocol procedure or study drug, the investigator should report the SAE to the sponsor, and the SAE will be entered in the Lilly Safety System.

Information on SAEs expected in the study population independent of drug exposure and that will be assessed by the sponsor in aggregate periodically during the course of the trial may be found in the IB

#### 10.3.1.2. Suspected Unexpected Serious Adverse Reactions

Suspected unexpected serious adverse reactions (SUSARs) are serious events that are not listed in the Development Core Safety Information in the IB and that the investigator identifies as related to the LY2835219 or study procedure. United States 21 CFR 312.32 and European Union Clinical Trial Directive 2001/20/EC and the associated detailed guidances or national regulatory requirements in participating countries require the reporting of SUSARs. Lilly has procedures that will be followed for the recording and expedited reporting of SUSARs that are consistent with global regulations and associated detailed guidances.

## 10.3.2. Other Safety Measures

#### 10.3.2.1. Electrocardiograms

For each patient receiving LY2835219, 12-lead digital ECGs will be collected according to the Study Schedule (Attachment 1) and Table JPBK.10.2 as single ECGs. For each patient receiving erlotinib, an ECG will be collected at baseline only. Patients must be supine for approximately 5 to 10 minutes before ECG collection and remain supine but awake during ECG collection.

 Table JPBK.10.2.
 Schedule for Electrocardiogram Collection

| Electrocardiogram | Cycle and Day | Timing |
|-------------------|---------------|------------------------------------------|
| 1 | Baseline | ≤14 Days |
| 2 | Cycle 1 Day 1 | Predose |
| 3 | Cycle 1 Day 1 | 4 to 6 hours postdose |
| 4 | Cycle 2 Day 1 | 4 to 6 hours postdose |
| 5 | Cycle 7 Day 1 | 4 to 6 hours postdose |
| 6 | Visit 801 | 30 days after study drug discontinuation |

Electrocardiograms may be obtained at additional times, when deemed clinically necessary. Collection of more ECGs than expected at a particular time point is allowed when needed to ensure high-quality records.

Electrocardiograms will be interpreted by a qualified physician (the investigator or qualified designee) at the site as soon after the time of ECG collection as possible, and ideally while the patient is still present, to determine whether the patient meets entry criteria and for immediate patient management, should any clinically relevant findings be identified.

After enrollment, if a clinically significant increase in the QT/QTc interval from baseline, or other clinically significant quantitative or qualitative change from baseline, is present, the investigator will assess the patient for symptoms (for example, palpitations, near syncope, or syncope) and to determine if the patient can continue in the study. The investigator or qualified designee is responsible for determining if any change in patient management is needed and must document his/her review of the ECG printed at the time of evaluation.

## 10.3.3. Safety Monitoring

The Lilly CRP will monitor safety data throughout the course of the study.

Lilly will review SAEs within time frames mandated by company procedures. The Lilly CRP will, as is appropriate, consult with the functionally independent GPS therapeutic area physician or clinical scientist, and review:

- trends in safety data
- laboratory analytes
- adverse events
- If a patient experiences elevated ALT >5× ULN and elevated total bilirubin >2× ULN, clinical and laboratory monitoring should be initiated by the investigator.
- Details for hepatic monitoring depend upon the severity and persistence of observed laboratory test abnormalities. To ensure patient safety and comply with regulatory guidance, the investigator is to consult with the Lilly CRP regarding collection of specific recommended clinical information and follow-up laboratory tests (see Attachment 3).

## 10.3.4. Complaint Handling

Lilly collects product complaints on study drugs used in clinical trials in order to ensure the safety of study participants, monitor quality, and to facilitate process and product improvements.

If supplied by Lilly, complaints related to unblinded comparator drugs are reported to Lilly. If sourced locally, complaints related to unblinded comparator drugs are reported directly to the manufacturers of those drugs in accordance with the package insert.

The investigator or his/her designee is responsible for handling the following aspects of the product complaint process in accordance with the instructions provided for this study:

- recording a complete description of the product complaint reported and any associated AEs using the study-specific complaint forms provided for this purpose
- faxing the completed product complaint form within 24 hours to Lilly or its designee

If the investigator is asked to return the product for investigation, he/she will return a copy of the product complaint form with the product.

## 10.4. Sample Collection and Testing

Attachment 1 lists the schedule for sample collections in this study.

Attachment 2 lists the specific tests that will be performed for this study and whether these will be performed at a central or local laboratory. Enrollment and treatment decisions may be based upon results of tests performed locally. If local laboratory tests are used for this purpose, then a duplicate specimen must be submitted to the central laboratory. Discrepancies between the local and central laboratory that may have an impact on eligibility or treatment decisions will not be considered protocol violations.

Attachment 6 provides a summary of the estimated maximum number and volume of invasive samples, for all sampling, during the study.

### 10.4.1. Samples for Study Qualification and Health Monitoring

Blood samples will be collected to determine whether patients meet inclusion/exclusion criteria and to monitor patient health.

Samples collected for specified laboratory tests will be destroyed within 60 days of receipt of confirmed test results. Tests are run and confirmed promptly whenever scientifically appropriate. When scientific circumstances warrant, however, it is acceptable to retain samples to batch the tests run, or to retain the samples until the end of the study to confirm that the results are valid. Certain samples may be retained for a longer period, if necessary, to comply with applicable laws, regulations, or laboratory certification standards.

## 10.4.2. Samples for KRAS Mutation Determination

To meet study eligibility criteria, and therefore mandatory for study participation, patients must have available FFPE tumor sample. While the tissue can be from either initial diagnosis or later (for example, at relapse), the most recent sample is preferred. The sample can be either 8 serially cut unstained sections (preferred) or a tissue block. Sample collection methods may include surgical resection, core needle biopsy, or fine needle aspirate. Due diligence should be used to make sure that tumor specimens (not a normal adjacent or a tumor margin sample) are provided.

*KRAS* mutation determination for study eligibility is made at the central laboratory using the QIAGEN<sup>®</sup> *therascreen*<sup>®</sup> KRAS RGQ PCR Kit NSCLC. Part of each patient's tumor tissue may be retained for repeat testing during the development of that investigational assay. The same sample used for *KRAS* mutant determination may also be used for evaluation of codons 12 and 13 via Sanger sequencing, and potentially an additional method, to test concordance with the investigational assay.

Prior local testing of *KRAS* status to informally assess eligibility for Study JPBK is highly discouraged. Submission of the investigational assay for potential regulatory approval requires a dataset containing evaluation of both *KRAS* mutant positive and negative samples. If local testing is completed per a site's standard of care, results should be disregarded when evaluating a patient's eligibility for the study.

Details for the handling and shipping of tumor biopsy samples will be provided in a separate document. Instructions and supplies required for the collection, processing, and shipment of the patients' samples will be provided by the sponsor.

The tumor tissue samples will be coded with the patient number and stored for up to a maximum 15 years after the last patient visit for the study at a facility selected by the sponsor. The samples and any data generated from them can only be linked back to the patient by investigator site personnel. The duration allows the sponsor to respond to regulatory requests related to the study drug. Tumor specimens submitted as a FFPE tissue block will be returned to the sites by end of study or upon request.

#### 10.4.3. Samples for Other Biomarkers

#### 10.4.3.1. Archived Tumor Tissue

An archived tumor sample will be collected on Cycle 1 Day 1 in addition to the sample used to determine *KRAS* mutation status. An FFPE tumor tissue sample OR 20 unstained slides are requested for further biomarker research. The tissue sample will be tested for biomarkers relevant to LY2835219 and the disease state and to correlate these markers to clinical outcome and to LY2835219. Analyses may include, but are not limited to, nucleic acid and protein profiles to better understand the disease process and to develop predictive biomarkers.

Any whole block submitted will be returned to the site. Any partial blocks or slides will either be returned or discarded within 15 years after last patient visit for the trial.

#### 10.4.3.2. Blood Samples for Pharmacogenetic Evaluations

There is growing evidence that genetic variation may impact a patient's response to therapy. Variable response to therapy may be due to genetic determinants that impact drug absorption, distribution, metabolism, and excretion, the mechanism of action of the drug, the disease etiology and/or the molecular subtype of the disease being treated. Therefore, where local regulations and ERBs allow, a blood sample will be collected for pharmacogenetic analysis.

Where local regulations and ERBs allow, a blood sample will be collected for pharmacogenetic analysis (refer to Attachment 1). Samples may be genotyped and analyses may be performed to evaluate a genetic association with response to LY2835219. These investigations may be limited to a focused candidate gene study or, if appropriate, genome-wide analysis may be performed to identify regions of the genome associated with the variability observed in drug response. The pharmacogenetic biomarker samples will only be used for investigations related to disease and drug or class of drugs under study in the context of this clinical program. They will not be used for broad exploratory unspecified disease or population genetic analysis.

The samples will be coded with the patient number and stored for up to a maximum 15 years after the last patient visit for the study at a facility selected by the sponsor. The samples and any data generated from them can only be linked back to the patient by investigator site personnel. The duration allows the sponsor to respond to regulatory requests related to the study drug.

Samples will be destroyed according to a process consistent with local regulation.

#### 10.4.3.3. Plasma Samples for Exploratory Biomarker Evaluations

Plasma samples will be collected and analysis may be performed on biomarkers that may play a role in the LY2835219 mechanism of action (refer to Attachment 1). The evaluation of these samples may involve analysis of DNA, RNA, and proteins (including any of these components derived from exosomes) to investigate their association with observed clinical outcomes to study drug. The samples will be coded with the patient number and stored for up to a maximum 15 years. Details for collecting, processing, and storing the samples are similar to those provided in Section 10.4.3.2.

## 10.4.4. Samples for Drug Concentration Measurements Pharmacokinetics

At the visits and times specified in the Pharmacokinetic Sampling Schedule (Attachment 7), 5 venous blood samples of approximately 2 mL each will be collected from patients receiving LY2835219 to determine the plasma concentrations of LY2835219 and its metabolites LSN2839567, LSN3106726, and LSN3106729. Patients receiving erlotinib will not have samples collected for PK analysis.

Separate blood samples are not required for the parent and its metabolites. Instructions for the collection and handling of blood samples will be provided by the sponsor. It is preferred that the blood samples be obtained from a peripheral location. Blood samples will be allowed from central access devices but a sample drawn from a central catheter of any type for PK must take precautions to prevent obtaining a dilute sample. If multiple samples are obtained centrally, the PK sample should be the last specimen drawn to reduce the potential for a diluted or improperly drawn sample. The actual date and time (24-hour clock time) of each sampling will be recorded. A maximum of 5 additional samples may be drawn at other time points during the study if warranted and agreed upon between both the investigator and Lilly.

These samples will be analyzed at a laboratory designated by the sponsor. Plasma concentrations of LY2835219 plus its metabolites LSN2839567, LSN3106726 and LSN3106729, will be assayed using a validated liquid chromatography/tandem mass spectrometry method. Bioanalytical samples collected to measure study drug concentration and metabolism and/or protein binding, will be retained for a maximum of 1 year following last patient visit for the study. The PK samples will be stored at a facility designated by the sponsor.

## 10.5. Appropriateness of Measurements

Efficacy measurements by radiographic imaging are standard, widely used, generally recognized as reliable, accurate, and able to discriminate between effective and ineffective agents.

Safety measurements by laboratory monitoring are standard, widely used, generally recognized as reliable, accurate, and able to discriminate between agents with acceptable and unacceptable safety profiles.

## 11. Data Quality Assurance

To ensure accurate, complete, and reliable data, Lilly or its representatives will do the following:

- provide instructional material to the study sites, as appropriate
- sponsor start-up training to instruct the investigators and study coordinators. This session will give instruction on the protocol, the completion of the CRFs, and study procedures.
- make periodic visits to the study site
- be available for consultation and stay in contact with the study site personnel by mail, telephone, and/or fax
- review and evaluate CRF data and use standard computer edits to detect errors in data collection
- conduct a quality review of the database

In addition, Lilly or its representatives will periodically check a sample of the patient data recorded against source documents at the study site. The study may be audited by Lilly or its representatives, and/or regulatory agencies at any time. Investigators will be given notice before an audit occurs.

To ensure the safety of participants in the study, and to ensure accurate, complete, and reliable data, the investigator will keep records of laboratory tests, clinical notes, and patient medical records in the patient files as original source documents for the study. If requested, the investigator will provide Lilly, applicable regulatory agencies, and applicable ERBs with direct access to original source documents.

## 11.1. Data Capture System

An electronic data capture system will be used in this trial. The site maintains a separate source for the data entered by the site into the sponsor-provided electronic data capture system.

Case report form data will be encoded and stored in a clinical trial database.

Any data for which the paper documentation provided by the patient will serve as the source document will be identified and documented by each site in that site's study file. Paper documentation provided by the patient may include, for example, a paper diary to collect patient-reported outcome measures (for example, a rating scale), a daily dosing schedule, or an event diary.

Data from complaint forms submitted to Lilly will be encoded and stored in the global product complaint management system.

## 12. Sample Size and Statistical Methods

## 12.1. Determination of Sample Size

The co-primary objectives of this study are to compare LY2835219 versus erlotinib with respect to PFS and OS in patients with Stage IV NSCLC whose tumors have detectable *KRAS* mutations (specifically, in codons 12 and 13 of the *KRAS* oncogene as determined by an investigational assay at the Study JPBK central laboratory) and who have progressed after prior platinum-based therapy and received 1 other prior therapy or are not eligible for further chemotherapy.

The study will enroll approximately 550 patients in 3:2 randomization (330 patients in the LY2835219 arm and 220 patients in the erlotinib arm). The primary PFS analysis will be performed after 338 PFS events have occurred. In order to ensure an adequate number of patients have been enrolled for the analysis of OS, the primary PFS analysis will not occur earlier than 2 months after the study enrollment is complete. The final OS analysis will occur when approximately 407 OS events have been observed.

Assuming a PFS HR of 0.67, this sample size yields approximately 80% statistical power to detect superiority of the LY2835219 arm over erlotinib arm with the use of a 2-sided log-rank test and a type I error of .005.

If the true median PFS for the erlotinib arm is 2 months, then the HR of 0.67 amounts to an approximately 1-month improvement in median PFS for the LY2835219 arm under an additional assumption of exponential survival distribution.

Assuming an OS HR of 0.75, this sample size yields approximately 80% statistical power to detect superiority of the LY2835219 arm over erlotinib arm with the use of a 2-sided log-rank test and a type I error of .045.

If the true median OS for the erlotinib arm is 6.5 months, then the HR of 0.75 amounts to an approximately 2.2-month improvement in median OS for the LY2835219 arm under an additional assumption of exponential survival distribution.

## 12.2. Statistical and Analytical Plans

#### 12.2.1. General Considerations

Statistical analysis of this study will be the responsibility of Lilly.

Efficacy analyses will be based on the intention-to-treat (ITT) analysis set. This population is defined as all patients randomized to study treatment. Patients will be grouped according to randomized treatment.

Safety analyses will be based on the Safety Population, defined as all enrolled patients receiving at least 1 dose of any study drug. Patients will be grouped according to treatment received in Cycle 1.

Pharmacodynamic and/or tailoring biomarker analyses will be based on the subset of patients from the above populations from whom a valid assay result (according to laboratory guideline) has been obtained.

All tests of treatment effects will be conducted at a 2-sided alpha level of 0.05, unless otherwise stated. All confidence intervals (CIs) will be given at a 2-sided 95% level, unless otherwise stated.

Any change to the data analysis methods described in the protocol will require an amendment ONLY if it changes a principal feature of the protocol.

Before unblinding of the aggregate database, minor modifications or clarifications to the data analysis methods may be described and justified in the statistical analysis plan (SAP).

Any other change to the data analysis methods described in the protocol, and the justification for making the change, will be described in the CSR.

The assumptions for each statistical method will be evaluated. If there is violation of assumptions, alternative statistical methods may be used.

Additional exploratory analyses of the data will be conducted as deemed appropriate.

#### 12.2.2. Patient Disposition

A detailed description of patient disposition will be provided. It will include a summary of the number and percentage of patients entered into the study, enrolled in the study, and treated as well as number and percentage of patients completing the study, or discontinuing (overall and by reason for discontinuation).

A summary of all important protocol deviations will be provided.

#### 12.2.3. Patient Characteristics

Patient demographics including age, sex, screening height and weight, screening body mass index, and smoking status will be reported using descriptive statistics.

Baseline disease characteristics will be summarized by presenting frequency counts and percentages for pathological diagnosis (histological or cytological), disease stage, or performance status.

Patient preexisting condition, historical illness, and prior chemotherapy (including both cytotoxic and targeted agents) will be summarized by treatment arm.

## 12.2.4. Concomitant Therapy

Concomitant medication will be summarized by treatment arm in a frequency table listing the terms recorded on the eCRF.

#### 12.2.4.1. Postdiscontinuation Therapy

The numbers and percentages of patients reporting postdiscontinuation therapies will be provided overall, by type of therapy (surgery, radiotherapy, or systemic therapy), and by drug name.

## 12.2.5. Treatment Compliance

The number of dose omissions, reductions, and delays, cycles received, and dose intensity will be summarized for all treated patients per treatment arm.

Treatment compliance information for LY2835219 or erlotinib will be collected through capsule (LY2835219) or tablet (erlotinib) counts at each tumor assessment visit. The estimate of percent compliance will be given by:

Percent Compliance = 
$$\frac{\text{Actual cumulative dose taken}}{\text{Expected cumulative dose to be taken}} \times 100$$

The actual cumulative dose taken will be determined based on counting the number of capsules returned at each visit and subtracting that number from the number of capsules dispensed. The expected cumulative dose to be taken will be determined based on the assigned dose and taking into account any dose reductions or omissions.

## 12.2.6. Primary Outcome and Methodology

The co-primary endpoints of this study are PFS and OS. The study-wise alpha of .05 will be split between the endpoints: .005 for PFS and .045 for OS. A fallback procedure will be used. The test on PFS will occur first; if the test on PFS is significant, the alpha used for this test will be added to the .045 originally allocated to OS for a total of .05. This fallback procedure will maintain a study-wise alpha level of .05. The alpha level used for each test at each analysis is described in Table JPBK.12.1.

Table JPBK.12.1. Alpha Allocation (2-Sided) for Progression-Free Survival and Overall Survival

| Endpoint | Alpha at PFS Analysis | Alpha at OS Analysis |
|---|---|---|
| | (338 PFS events) | (407 OS events) |
| PFS | .005 | |
| OS (If PFS is significant) | .001 | .049 |
| OS (If PFS is not significant) | .001 | .044 |

Abbreviations: OS = overall survival; PFS = progression-free survival.

PFS time is measured from the date of randomization to the date of investigator-determined objective progression as defined by RECIST v1.1, or death from any cause. Patients who have neither progressed nor died will be censored at the day of their last radiographic tumor assessment (if available) or date of randomization if no post initiation (that is, postbaseline) radiographic assessment is available. All randomized patients, according to the ITT principle,

will be included in the analysis of both endpoints. The detailed censoring rules for PFS are described in Table JPBK.12.2.

Table JPBK.12.2. Rules for Determining Date of Progression or Censor for Progression-Free Survival

| | Situation | Date of Progression or Censor | Outcome |
|---|---|---|---|
| 1 | No baseline tumor assessments | Date of Randomization | Censored |
| 2 | No post baseline assessments and no death | Date of Randomization | Censored |
| 3 | No documented progression and no death (with a post-baseline tumor assessment) | Date of last adequate tumor assessment | Censored |
| 4 | Patient lost to follow-up (or withdrew consent<br>from study participation) before documented<br>progression or death | Date of last adequate tumor assessment | Censored |
| 5 | Documented progression | Date of documented progression. If a tumor assessment was done on multiple days, use the earliest date for that visit. | Progressed |
| 6 | Death without documented progression | Date of death | Progressed |
| 7 | Death or documented progression immediately after missed ≥2 consecutive post-baseline tumor assessment visits | Date of last adequate tumor assessment<br>before missed assessments or date of<br>randomization, whichever is later | Censored |

Note: Progression-free survival and associated outcome is determined by the earliest of the dates above, if more than 1 situation applies.

Overall survival duration is measured from the date of randomization to the date of death from any cause. For each patient who is not known to have died as of the data-inclusion cutoff date for a particular analysis, OS will be censored for that analysis at the date of last contact prior to the data inclusion cutoff date (contacts considered in the determination of last contact date include AE date, lesion assessment date, visit date, and last known alive date).

The comparison of each of the PFS and OS distributions between treatment groups will be conducted using a stratified log-rank test with the following stratification variables: number of prior chemotherapy regimens (1 versus 2), ECOG PS (0 versus 1), gender (male versus female), and KRAS mutation (G12C versus all others).

The Kaplan-Meier method (Kaplan and Meier 1958) will be used to estimate the PFS and OS survival curves as well as survival rates at 3, 6, 9, and 12 months for each treatment group. These rates will be compared based on a normal approximation for the difference between the rates.

The Cox proportional hazard model (Cox 1972) with treatment as a factor, stratified by the stratification factors used in the randomization (as per the primary analysis) will be used to estimate the HR and corresponding 95% CI.

## 12.2.7. Secondary Outcome and Methodology

The secondary objectives for this study are stated in Section 6.2.

The objective response rate of each treatment arm will be calculated as defined by RECIST v1.1. All rates will be compared between treatment arms based on a normal approximation for the difference between the rates.

## 12.2.8. Sensitivity Analysis

Sensitivity analyses will be undertaken for calculation of the primary endpoint in order to evaluate the robustness of the analysis. The following sensitivity analyses will be performed for PFS:

**Progression-Free Survival Sensitivity Analysis 1** (censoring for receiving subsequent systemic anticancer therapy): if a patient is initiated on another anticancer therapy prior to objective progression, including any postdiscontinuation treatment systemic therapy, radiotherapy, or surgical intervention, PFS will be censored at the date of the last complete objective progression-free disease assessment before initiation of the new therapy, regardless of whether or not this patient subsequently had objective progression or died.

**Progression-Free Survival Sensitivity Analysis 2** (nonobjective progression as a PFS event): if a patient is discontinued from study treatment due to investigator determined non-objective progression (for example, symptomatic deterioration), then the patient's PFS time will be calculated using the date of non-objective progression as the progression date.

**Progression-Free Survival Sensitivity Analysis 3** (back-dating progressions at unscheduled assessments): if a patient has objective progression at an unscheduled disease assessment, then the PFS time for that patient will be back-dated to the prior scheduled disease assessment.

## 12.2.9. Pharmacokinetic Analyses

Pharmacokinetics analyses will be conducted on all patients who have received at least 1 dose of LY2835219 and have had samples collected (see PK sampling schedule in Attachment 7).

Mean population PK parameters for LY2835219 in plasma (clearance, exposure, volume of distribution, and half-lives) and inter-individual PK variability will be computed using nonlinear mixed effect modeling (NONMEM). The current PK model for LY2835219, which has been developed using plasma concentration data available from the Phase 1 Study JPBA, will be updated using the plasma data collected in this study. Covariate effects (such as age, weight, sex, creatinine clearance, and plasma protein levels) on the PK parameters of LY2835219 in plasma will also be investigated.

The mean population PK properties of LY2835219 metabolites LSN2839567, LSN3106726, and LSN3106729 in plasma may also be analyzed by means of NONMEM.

Finally, pharmacodynamic data (such as neutrophil, lymphocytes, or platelets counts in blood) collected in this study may also be analyzed by means of NONMEM and connected to the population PK model in a PK/pharmacodynamic model.

The version of software used for the analysis will be documented and will meet the Lilly requirements of software validation.

### 12.2.10. Biomarker Analyses

#### 12.2.10.1. KRAS Mutation Assessment

Concordance (agreement) analysis will be performed on samples with valid *KRAS* status (mutation positive and mutation negative) using both the investigational assay and the reference method (Sanger sequencing). Measures of agreement between the investigational *KRAS* assay and the reference method, including positive percent agreement, negative percent agreement, and overall percent agreement, and their corresponding exact 2-sided 95% CIs, will be estimated for the overall mutation status; that is, mutation detected or not detected for the 7 mutations of *KRAS* gene. A secondary agreement analysis between the investigational *KRAS* assay and the reference method will be performed for each of the tumor tissue sample types (surgical resection, fine needle aspirate and core needle biopsy). The data will also be summarized for each of the 7 *KRAS* mutations separately.

#### 12.2.10.2. Other Biomarkers

For other biomarkers relevant to LY2835219 and the disease state, the distributions of biomarkers will be summarized for the patient population for which samples are available. Associations between clinical endpoints and biomarkers will be evaluated using data from patients who have an evaluable sample for each biomarker of interest, and such evaluation will be done on an individual marker basis.

#### 12.2.11. Health Outcome/Quality of Life Analyses

Patient-reported outcomes are measured through paper versions of the following:

- MDASI-LC (includes additional page with 11 items that will be scored separately)
- EQ-5D 5L (EuroQol 5-Dimension 5 Level)

The reason and number of missing and incomplete questionnaires/assessments by visit will be summarized for each instrument and study arm.

#### 12.2.11.1. MDASI-LC

The MDASI-LC population will include all patients who completed at least 1 baseline followed by at least 1 MDASI-LC assessment after 1 cycle of study drug (Cycle 2 Day 1 or later).

The MDASI-LC will be summarized for each assessment period and scored as described (Mendoza et al. 2011). The instrument will be reported as core symptoms (Items 1-13), interference items (Items 14-19) and lung symptoms (Items 14-16), and the 11 additional items will be reported as brain tumor symptoms (Items 23 through 30) and additional 3 items (31-33), as well as each individual item.

For each patient with data from baseline and at least 1 other visit, the maximum change from baseline score will be calculated and summarized for MDASI-LC composite scores, and "worst pain".

Further analysis details will be described in the SAP.

#### 12.2.11.2. Health State Utility

The EQ-5D 5L population will include all patients who completed at least 1 baseline followed by at least 1 EQ-5D 5L assessment after 1 dose of study drug.

The EQ-5D 5L data will be scored based on EuroQol recommendations. The index score is calculated from a set of item weights to derive a score of <0 to 1, with 1 representing the best health status. The visual analogue score (VAS) is scored from 0 (worst imaginable health state) through 100 (best imaginable health state) to represent the patient's self-report for each day. EQ-5D 5L responses for each item will be summarized by frequency and corresponding percentages. Descriptive statistics for the index and VAS will be calculated as described in the SAP.

#### 12.2.11.3. Use of Pain Medications

Pain medication will be classified into 1 of 6 categories by the sponsor, using an analgesic ladder approach with medication category based on a World Health Organization scale outlined in Table JPBK.12.3. A therapy category for each cycle will be assigned according to the maximum category of therapy administered based on analgesic data from the Concomitant Form for that cycle. Category of pain medication for each cycle will be determined based on the data collected on analgesic use by Anatomical Therapeutic Chemical code. Change in categories based on analgesic ladder compared to baseline will be described by arm.

 Table JPBK.12.3.
 World Health Organization Pain Scale

| Code | Description |
|---|---|
| 0 | No analgesia |
| 1 | Aspirin (for pain, not cardiovascular prophylaxis), acetaminophen, nonsteroidal anti-inflammatory drugs |
| 2 | Codeine, hydrocodone, pentazocine, oxycodone |
| 3 | Oral morphine, hydromorphone, methadone, transdermal fentanyl |
| 4 | Parenteral opiates |
| 5 | Neurosurgical procedures (blocks) |

## 12.2.12. Safety Analyses

All safety summaries and analyses will be based upon the Safety Population as defined in Section 12.2.1.

Overall exposure to study drug, the numbers of patients completing each cycle, and the dose intensity will be summarized using descriptive statistics. The number of patients with dose reductions, dose delays, or dose omissions will also be summarized, as will the reasons for dose adjustments.

AEs will be reported using a unified CTCAE/MedDRA reporting process:

- The CTCAE v4.03 term reported by the investigator will be mapped to the MedDRA Preferred Term (PT) and System Organ Class (SOC) of the corresponding MedDRA Lower Level Term (LLT), unless the reported CTCAE term is 'Other specify'.
- If the reported CTCAE term is 'Other specify' the MedDRA LLT, PT, and SOC mapped from the verbatim AE term will be used.

• All listings and summaries will use the PT resulting from this process.

Preexisting conditions are defined as adverse events that begin prior to the first dose of study drug. A treatment-emergent adverse event (TEAE) is defined as an event that first occurred or worsened in severity after baseline. Comparisons of preexisting conditions to on-treatment events at the LLT level will be used in the treatment-emergent computation.

An overall summary of AEs will be provided for AEs deemed by the investigator to be possibly related to study drug, and repeated for events regardless of study drug causality. Incidence rates of these events will be compared between treatment arms using Chi square test.

The following summaries will be produced by PT within SOC: preexisting conditions, SAEs, TEAEs, drug-related TEAEs, and procedure-related TEAEs.

The following summaries will be produced by PT within SOC and maximum CTCAE grade: laboratory-based TEAEs, nonlaboratory-based TEAEs, drug-related laboratory-based TEAEs, and drug-related nonlaboratory-based TEAEs.

Reasons for death will be summarized separately for on-therapy and within 30 days of treatment discontinuation.

Hospitalizations and transfusions during the study treatment period or during the 30-day short-term follow-up period will be summarized by treatment group.

## 12.2.13. Subgroup Analyses

Subgroup analyses of PFS and OS will be performed for potential prognostic and predictive subgroup variables.

## 12.2.14. Interim Analyses

## 12.2.14.1. Safety Interim Analyses

The data monitoring committee (DMC) is responsible for providing external oversight of patient safety in Study JPBK independently of the Lilly study team and Lilly GPS.

During the study, safety interim analyses will be performed approximately every 6 months. The safety interim analyses will be conducted to evaluate the overall safety profile of LY2835219. At the recommendation of the DMC, the frequency of safety interim analyses may be modified.

At each interim analysis, the DMC may recommend the trial continue without modifications, continue with specific modifications, or be stopped for safety concerns. There will be no prespecified rules for stopping the trial due to safety concerns. The DMC members will review unblinded safety data at each interim analysis. If a significant safety signal is identified, the DMC may recommend a protocol amendment, termination of enrollment, and/or termination of study treatment. The recommendations of the DMC will be communicated to the Lilly Senior Management Designee and, if necessary, an Internal Review Committee.

In the event that safety monitoring uncovers an issue that needs to be addressed by unblinding at the treatment group level, members of the DMC can conduct additional analyses of the safety

data. Additionally, unblinding of a limited number of Lilly representatives external to the study team may be required for evaluation of selected SAEs for determination of regulatory reporting.

### 12.2.14.2. Efficacy Interim Analyses

One interim futility analysis will be performed by an independent DMC. The analysis will occur after 100 PFS events have been observed. The DMC will be instructed to recommend the study be stopped for futility if the observed hazard ratio for PFS (as calculated using a stratified Cox proportional hazards model) is greater than 0.95.

Only the DMC is authorized to evaluate unblinded interim efficacy and safety analyses. Study sites will receive information about interim results ONLY if they need to know for the safety of their patients.

## 13. Informed Consent, Ethical Review, and Regulatory Considerations

#### 13.1. Informed Consent

The investigator is responsible for ensuring that the patient understands the potential risks and benefits of participating in the study, including answering any questions the patient may have throughout the study and sharing in a timely manner any new information that may be relevant to the patient's willingness to continue his or her participation in the trial.

There may be 2 ICF used in this study: pre-screening ICF and study ICF.

The pre-screening ICF will provide relevant information and to document that the patient is satisfied with his or her understanding of the genetic testing of the tumor sample for *KRAS* mutation status. No procedures will be conducted or treatment provided to patients after signing this pre-screening ICF. Pre-screening is optional; the determination may also be made during screening under the study ICF.

The study ICF will be used to explain the potential risks and benefits of study participation to the patient in simple terms before the patient is entered into the study, and to document that the patient is satisfied with his or her understanding of the risks and benefits of participating in the study and desires to participate in the study. If determination of *KRAS* mutation status by the Study JPBK central laboratory was not completed during a pre-screening period, then the determination will be made during screening under the study ICF.

The investigator is responsible for ensuring that informed consent is given by each patient or legal representative. This includes obtaining the appropriate signatures and dates on the ICF prior to the performance of any protocol procedures and prior to the administration of study drug.

As used in this protocol, the term "informed consent" includes all consent and assent given by patients or their legal representatives.

#### 13.2. Ethical Review

Lilly or its representatives must approve all ICFs before they are used at the investigative sites. All ICFs must be compliant with the International Conference on Harmonisation (ICH) guideline on GCP.

Documentation of ERB approval of the protocol and the ICF must be provided to Lilly before the study may begin at the investigative sites.

The study site's ERBs should be provided with the following:

- the current IB or package labeling (for example, PI or SmPC) and updates during the course of the study
- ICF
- relevant curricula vitae

#### 13.3. Regulatory Considerations

This study will be conducted in accordance with:

- consensus ethics principles derived from international ethics guidelines, including the Declaration of Helsinki and Council for International Organizations of Medical Sciences International Ethical Guidelines
- the ICH GCP Guideline (E6)
- applicable laws and regulations.

The investigator or designee will promptly submit the protocol to applicable ERB(s).

Some of the obligations of Lilly will be assigned to a third-party organization.

An identification code assigned to each patient will be used in lieu of the patient's name to protect the patient's identity when reporting AEs and/or other trial-related data.

## 13.3.1. Investigator Information

Physicians with a specialty in oncology will participate as investigators in this clinical trial.

## 13.3.2. Protocol Signatures

The sponsor's responsible medical officer will approve the protocol, confirming that, to the best of his or her knowledge, the protocol accurately describes the planned design and conduct of the study.

After reading the protocol, each principal investigator will sign the protocol signature page and send a copy of the signed page to a Lilly representative.

## 13.3.3. Final Report Signature

The clinical study report (CSR) coordinating investigator will sign the final CSR for this study, indicating agreement that, to the best of his or her knowledge, the report accurately describes the conduct and results of the study.

Lilly will select an investigator to serve as the CSR coordinating investigator.

The Lilly responsible medical officer and statistician will sign/approve the final CSR for this study, confirming that, to the best of his or her knowledge, the report accurately describes the conduct and results of the study.

#### 14. References

- Brugger W, Triller N, Blasinska-Morawiec M, Curescu S, Sakalauskas R, Manikhas GM, Mazieres J, Whittom R, Ward C, Mayne K, Trunzer K, Cappuzzo F. Prospective molecular marker analyses of EGFR and KRAS from a randomized, placebo-controlled study of erlotinib maintenance therapy in advanced non-small-cell lung cancer. *J Clin Oncol*. 2011;29(31):4113-4120.
- Cancer Therapy Evaluation Program, Common Terminology Criteria for Adverse Events, Version 4.0, DCTD, NCI, NIH, DHHS. 2009. Publish date: 29 May 2009.
- Ciuleanu T, Stelmakh L, Cicenas S, Miliauskas S,Grigorescu AC, Hillenbach C, Johannsdottir HK, Klughammer B, Gonzalez EE. Efficacy and safety of erlotinib versus chemotherapy in second-line treatment of patients with advanced, non-small-cell lung cancer with poor prognosis (TITAN): a randomised multicentre, open-label, phase 3 study. *Lancet Oncol.* 2012;13(3):300-308.
- Cox DR. Regression models and life-tables. J Royal Stat Soc Ser B. 1972;74(2):187-220.
- Edge SB, Byrd DR, Compton CC, Fritz AG, Greene FL, Trotti A, eds. AJCC Cancer Staging Handbook: From the AJCC Cancer Staging Manual. 7th ed. NY: Springer; 2009.
- Eisenhauer EA, Therasse P, Bogaert J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). *Eur J Cancer*. 2009;45(2):228-247.
- [FDA] US Food and Drug Administration. Information on Erythropoiesis Stimulating Agents. Available at: http://www.fda.gov/Drugs/DrugSafety/PostmarketDrugSafety InformationforPatientsandProviders/UCM109375. Accessed 28 July 2009.
- Garassino MC, Martelli O, Broggini M, Farina G, Veronese S, Rulli E, Bianchi F, Bettini A, Longo F, Moscetti L, Tomirotti M, Marabese M, Ganzinelli M, Lauricella C, Labianca R, Floriani I, Giaccone G, Torri V, Scanni A, Marsoni S; TAILOR trialists. Erlotinib versus docetaxel as second-line treatment of patients with advanced non-small-cell lung cancer and wild-type EGFR tumours (TAILOR): a randomised controlled trial. *Lancet Oncol*. 2013;14(10):981-988.
- Gralla RJ, Roila F, Tonato M, Herrstedt J (Organizing and Overall Meeting Chairs). Multinational Association of Supportive Care in Cancer Consensus Conference on Antiemetic Therapy, Latest Update: April 2010. Available at: http://www.mascc.org/.
- Guan JL, Zhong WZ, An SJ, Yang JJ, Su J, Chen ZH, Yan HH, Chen ZY, Huang ZM, Zhang XC, Nie Q, Wu YL. KRAS mutation in patients with lung cancer: a predictor for poor prognosis but not for EGFR-TKIs or chemotherapy. *Ann Surg Oncol*. 2013;20(4):1381-1388.
- Janssen MF, Birnie E, Haagsma JA, Bonsel GJ. Comparing the standard EQ-5D three-level system with a five-level version. *Value in Health*. 2008;11(2):274-284.
- Kaplan EL, Meier P. Nonparametric estimation of incomplete observations. *J Amer Stat Assoc.* 1958;53:457-481.

- Kris MG, Hesketh PJ, Somerfield MR, Feyer P, Clark-Snow R, Koeller JM, Morrow GR, Chinnery LW, Chesney MJ, Gralla RJ, Grunberg SM; American Society of Clinical Oncology. American Society of Clinical Oncology guideline for antiemetics in oncology: update 2006. *J Clin Oncol*. 2006;24(18):2932-2947.
- Langer CJ. Roles of EGFR and KRAS Mutations in the treatment of patients with non-small-cell lung cancer. *Pharmacy Therapeutics*. 2011;36(5):263-268, 277-279.
- Linardou H, Dahabreh IJ, Kanaloupiti D, Siannis F, Bafaloukos D, Kosmidis P, Papadimitriou CA, Murray S. Assessment of somatic k-RAS mutations as a mechanism associated with resistance to EGFR-targeted agents: a systematic review and meta-analysis of studies in advanced non-small-cell lung cancer and metastatic colorectal cancer. *Lancet Oncol.* 2008;9(10):962-972.
- Mendoza TR, Wang XS, Lu C, Palos GR, Liao Z, Mobley GM, Kapoor S, Cleeland CS. Measuring the symptom burden of lung cancer: the validity and utility of the lung cancer module of the M. D. Anderson Symptom Inventory. *Oncologist*. 2011;16(2): 217-227.
- Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the eastern cooperative oncology group. *Am J Clin Oncol*. 1982;5:649-655.
- Puyol M, Martin A, Dubus P, Mulero F, Pizcueta P, Khan G, Guerra C, Santamaría D, Barbacid M. A synthetic lethal interaction between K-Ras oncogenes and Cdk4 unveils a therapeutic strategy for non-small cell lung cancer. *Cancer Cell*. 2010;18(1): 63-73.
- Rizzo JD, Somerfield MR, Hagerty KL, Seidenfeld J, Bohlius J, Bennett CL, Cella DF, Djulbegovic B, Goode MJ, Jakubowski AA, Rarick MU, Regan DH, Lichtin AE; American Society of Clinical Oncology; American Society of Hematology. Use of epoetin and darbepoetin in patients with cancer: 2007 American Society of Clinical Oncology/American Society of Hematology clinical practice guideline update. *J Clin Oncol.* 2008;26(1):132-149. Erratum in: *J Clin Oncol.* 2008;26(7):1192.
- Tarceva [US package insert]. Melville, NY: OSI Pharmaceuticals, Inc.; 2010. Available at: www.accessdata.fda.gov/drugsatfda\_docs/label/2010/021743s14s16lbl.pdf. Accessed April 15, 2014.
- Zhu CQ, da Cunha Santos G, Ding K, Sakurada A, Cutz JC, Liu N, Zhan T, Marrano P, Whitehead M, Squire JA, Kamel-Reid S, Seymour L, Shepherd FA, Tsao MS. Role of *KRAS* and *EGFR* as biomarkers of response to erlotinib in National Cancer Institut of Canada Clinical Trials Group Study BR.21. *J Clin Oncol* 2008;26(26):4268-4275.

## Attachment 1. Protocol JPBK Study Schedule

## Study Schedule, Protocol I3Y-MC-JPBK

Perform procedure as indicated.

| | | | Pre-<br>Screen <sup>a</sup> | Baseline | | Patients on Study Treatment | | | Postdiscontinuation<br>Follow-Up | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Cycle | Pre-<br>screening<br>BL | I | BL | 1 | 2 | 3 – n | Short-<br>Term<br>Follow-<br>Upb | Long-<br>Term<br>Follow-<br>Up |
| | | Visit | PRE0 | | 0 | 1 | 2 | 3 – n | 801 | 802 -<br>8XX |
| | | Duration (days) | | <u> </u> | 28 | 28 | 28 | 28 | 30 | 60 |
| | | Relative<br>day within<br>a cycle | | ≤28 | ≤14 | 1 | 1 | 1 | | |
| Procedure<br>Category | Procedure | Protocol<br>Reference | | | | | | | | |
| Study Entry<br>/Enrollment | Informed Consent<br>Form signed (prior to<br>performance of any<br>protocol-specific<br>tests/procedures) | Section<br>13.1 | Х | | X | | | | | |
| /Enronment | Inclusion/Exclusion evaluation | Section 7 | X | X | | | | | | |
| | Brain scan <sup>c</sup> | Section 7.1 | | X | | | | | | |
| | Initial history/<br>preexisting conditions | | | | X | | | | | |
| Medical<br>History | Historical illnesses | | | | X | | | | | |
| | Smoking/alcohol habits assessment | | | | X | | | | | |
| | Height | | | | X | | | | | |
| | Weight | | | | X | | X | X | X | |
| Physical<br>Examination | Blood pressure/pulse | Section 10.3.1 | | | X | | X | X | X | |
| | ECOG performance status | Section<br>Attachment<br>4 | | | X | X | X | X | X | |
| | Tumor measurement (palpable or visible) <sup>d</sup> | Section<br>10.1 | | | X | | X | X | | Xe |
| Tumor<br>Assessment | Radiologic imaging according to RECIST f | Section<br>10.1<br>Attachment<br>5 | | | X | | | Х | X | Xe |
| Survival infor | mation | Section<br>10.1 | | | | | | | X | Xg |
| Adverse Event<br>Gradingh | : Collection/CTCAE | Section<br>10.3 | | | X | X | X | X | X | X |

| | | | Pre-<br>Screen <sup>a</sup> | Baseline | | Patients on Study Treatment | | eatment | Postdiscontinuation<br>Follow-Up | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Cycle | Pre-<br>screening<br>BL | В | L | 1 | 2 | 3 – n | Short-<br>Term<br>Follow-<br>Upb | Long<br>Term<br>Follow-<br>Up |
| | | Visit | PRE0 | ( | ) | 1 | 2 | 3 – n | 801 | 802 -<br>8XX |
| | | Duration (days) | | ≤. | 28 | 28 | 28 | 28 | 30 | 60 |
| | | Relative day within a cycle | | ≤28 | ≤14 | 1 | 1 | 1 | | |
| Procedure<br>Category | Procedure | Protocol<br>Reference | | | | | | | | |
| Concomitant N | Medication Notation | Section 9.6 | | | X | X | X | X | X | |
| | Central hematology i | Section Attachment 2 | | | X | X | X | X | X | |
| | Central chemistry i | Section Attachment 2 | | | X | X | X | X | X | |
| | Local serum pregnancy test j | Section Attachment 2 | | | X | | χk | χk | | |
| Lab/<br>Diagnostic | Central pharmacokinetic sampling <sup>1</sup> | Section<br>Attachment 7 | | | | X | X | X | | |
| Tests | Pharmacogenetic blood sample | Section 10.4.3.2 | | | | X | | | | |
| | Plasma sample for circulating biomarkers | Section 10.4.3.3 | | | | X | X m | | | |
| | Local ECG n | Section 10.3.2.1 | | | хо | хр | χq | Хr | X s | |
| | Archived tumor samples | Section 10.4.2<br>and 10.4.3.1 | X t | χu | | χv | | | | |
| Health | MDASI-LC W | Section 10.2 | | | X | | X | X | X | |
| Outcomes<br>Assessments | EQ-5D 5L w | Section 10.2 | | | X | | X | X | X | |
| Study Drug | LY2835219 X | Section 9.1 | | | | X | X | X | | |
| Study Drug | Erlotinib Y | Section 9.1 | | | | X | X | X | | |

Abbreviations: BL = baseline; CNS = central nervous system; CTCAE = Common Terminology Criteria for Adverse Events; ECG = electrocardiogram; ECOG = Eastern Cooperative Oncology Group; EQ-5D 5L = European Quality of Life – 5 Dimensions – 5 Level; FFPE = formalin-fixed paraffin-embedded; ICF = informed consent form; MDASI-LC = MD Anderson Symptom Inventory; MRI = magnetic resonance imaging; OS = overall survival; PK = pharmacokinetics; RECIST = Response Evaluation Criteria in Solid Tumors; SAEs = serious adverse events; V = Visit.

- <sup>a</sup> The pre-screening period begins when the pre-screening ICF is signed for evaluation of FFPE tissue and ends once the *KRAS* mutation status of the tissue is determined. This period is optional; *KRAS* mutation status can also be determined during screening under the study ICF.
- b Short-term follow up begins the day after the patient and the investigator agree that the patient will no longer continue study treatment and lasts approximately 30 days.
- c Patients with a history of CNS metastases must have a brain scan (for example, MRI) within 28 days of randomization to document stability of their CNS metastases, even if there have been no changes in symptoms.

#### Study Schedule, Protocol I3Y-MC-JPBK (concluded)

- d Palpable or visual tumor measurement to be performed within 72 hours of start of each cycle if assessed as target/non-target lesions.
- e For patients who discontinue study treatment without objectively measured progressive disease, continue to evaluate tumor response every 8 weeks by the same method used at baseline and throughout the study until the patient has objective disease progression, or until the study's final analysis of OS. After the patient has objective disease progression, radiologic tests are no longer required and the patient will be followed up approximately every 60 days (±14 days) until the patient's death or overall study completion.
- f Imaging studies are performed locally and transmitted for central review. Radiological assessment of the chest and abdominal region is performed at baseline (Day -28 to Day-1), then on Day 1 (or up to 7 days before Day 1) of every other cycle beginning with Cycle 3 until progressive disease or start next line of anti-tumor treatment. If a cycle is delayed, tumor assessment should be concurrent with Day 1 of the new cycle.
- g Collection of survival data and subsequent antitumor therapies. Every 60 days (±14 days). Whenever possible, survival follow-up is conducted in person. If an in-person visit is not possible, the site may confirm survival by contacting the patient directly via phone.
- Data on SAEs that occur before the end of trial will be stored in the collection database and the Lilly Safety System. During long-term follow-up, only SAEs that are related to protocol procedures or study drug will be collected. All drug- or procedure-related adverse events and serious adverse events should be followed until they resolve, are no longer considered to be drug- or procedure-related, become stable or return to baseline, the patient starts a new therapy, the patient dies, or the patient becomes lost to follow-up. Frequency of evaluation is left to the judgment of the investigator.
- i Laboratory assessments should occur on Day 1 (±3 days) of the cycle. If the baseline laboratory assessment was conducted ≤3 days prior to Cycle 1 Day 1, reassessment is not required at Cycle 1 Day 1. For central versus local labs, refer to Attachment 2.
- j Perform pregnancy tests for woman of child-bearing potential.
- k Perform pregnancy tests once every 28 days (±7 days) prior to administration of study drug, where required by local regulations.
- 1 Sparse PK samples will be collected on Cycle 1 Day 1, Cycle 2 Day 1 and Cycle 3 Day 1.
- m This plasma sample should be collected on Cycle 2 Day 1.
- n Local ECG (no replicates required).
- o A baseline ECG will be collected from all patients.
- P ECG will be collected from patients receiving LY2835219 only. Two ECG will be collected on Cycle 1 Day 1. The first ECG will be collected predose; the second will be collected 4 to 6 hours postdose.
- 9 ECG will be collected from patients receiving LY2835219 only. An ECG will be collected 4 to 6 hours postdose on Cycle 2 Day 1.
- <sup>r</sup> If the patient received LY2835219 for 6 months, an additional ECG will be collected 4 to 6 hours postdose Cycle 7 Day 1.
- s ECG will be collected from patients receiving LY2835219 only.
- t Formalin-fixed paraffin-embedded tumor tissue requested after patient signs pre-screening ICF. Eight slides are mandatory for *KRAS* testing by the Study JPBK central laboratory prior to enrollment. If testing did not occur during pre-screening, sample collection and testing is required during baseline visit.
- <sup>u</sup> If the patient was not pre-screened, FFPE tumor tissue requested after patient signs the study ICF. Eight slides are mandatory for *KRAS* testing by the Study JPBK central laboratory prior to enrollment.
- v An additional 20 slides or FFPE tumor tissue block requested for biomarker research.
- w MDASI-LC and EQ-5D 5L should be administered at baseline (Day-14 to Day -1), on Day 1 of every cycle beginning with Cycle 2, and at the 30-day follow up visit (V801). The preferred order of collection is MDASI-LC and then EQ-5D 5L. Patients should complete before interaction with site staff.
- x LY2835219 is to be administered every 12 hours (± approximately 2 hours) on Days 1 through 28 of each cycle.
- Erlotinib is to be administered every 24 hours (± approximately 2 hours) on Days 1 through 28 of each cycle.

#### Study Schedule for the extension period only, Protocol I3Y-MC-JPBK]

Patients receiving LY2835219 and experiencing ongoing clinical benefit may continue to receive LY2835219 in the extension period. Patients receiving erlotinib will be discontinued from the study and cross-over to LY2835219 is not allowed.

Perform procedure as indicated.

| | | | Patients on Study Treatment | Extension Period Follow-Up |
|---|---|---|---|---|
| | | Cycle | 2-n | Follow-Up <sup>a</sup> |
| | | Visit | 501-5XX | 901 |
| | | Duration (days) | 28 | 30 |
| | | Relative day<br>within a<br>cycle | 1 | |
| Procedure<br>Category | Procedure | Protocol<br>Reference | | |
| Adverse Even<br>Grading <sup>b</sup> | ts Collection/CTCAE | Section<br>10.3.1 | X | X |
| Study Drug | LY2835219 <sup>c</sup> | Section 9.1 | X | |

Abbreviations: CTCAE = Common Terminology Criteria for Adverse Events; PK = pharmacokinetics; SAEs = serious adverse events.

- a The extension period begins after study completion and ends at the end of trial.
- b Data on SAEs that occur before the end of trial will be stored in the collection database and the Lilly safety system.
- <sup>c</sup> LY2835219 is to be administered every 12 hours (± approximately 2 hours) on Days 1 through 28 of each cycle. Note: Efficacy assessments will be done at the investigator's discretion based on the standard of care.

## **Attachment 2. Protocol JPBK Clinical Laboratory Tests**

#### **Clinical Laboratory Tests**

HematologyaClinical ChemistryaHemoglobinSerum Concentrations of:

Hematocrit Sodium

Erythrocyte count (RBC) Potassium

Mean cell volume (MCV) Chloride

Mean cell hemoglobin concentration (MCHC) Total bilirubin

Leukocytes (WBC) Direct bilirubin

Neutrophils Alkaline phosphatase

LymphocytesAlanine aminotransferase (ALT)MonocytesAspartate aminotransferase (AST)EosinophilsBlood urea nitrogen (BUN)

Basophils Creatinine
Platelets Calcium
Albumin
Total Protein

Pregnancy Test (females only)b

Serum

Abbreviations: RBC = red blood cells; WBC = white blood cells.

- a Assayed by Lilly-designated laboratory.
- b Local or investigator-designated laboratory.

#### Other Laboratory Tests<sup>a</sup>

KRAS

Sanger Sequencing

<sup>&</sup>lt;sup>a</sup> Assayed by Lilly-designated laboratory.

## Attachment 3. Protocol JPBK Hepatic Monitoring Tests for Treatment-Emergent Abnormality

Selected tests may be obtained in the event of a treatment-emergent hepatic abnormality and may be required in follow up with patients in consultation with the Lilly clinical research physician.

| Hepatic Hematologya | Haptoglobin <sup>a</sup> |
|------------------------|-----------------------------------|
| Hemoglobin | Tuptogroom |
| Hematocrit | Hepatic Coagulationa |
| RBC | Prothrombin Time |
| WBC | Prothrombin Time, INR |
| Neutrophils, segmented | |
| Lymphocytes | Hepatic Serologies <sup>a,b</sup> |
| Monocytes | Hepatitis A antibody, total |
| Eosinophils | Hepatitis A antibody, IgM |
| Basophils | Hepatitis B surface antigen |
| Platelets | Hepatitis B surface antibody |
| | Hepatitis B Core antibody |
| Hepatic Chemistrya | Hepatitis C antibody |
| Total bilirubin | Hepatitis E antibody, IgG |
| Direct bilirubin | Hepatitis E antibody, IgM |
| Alkaline phosphatase | 1 |
| ALT | Anti-nuclear antibodya |
| AST | · |
| GGT | Anti-smooth muscle antibodya |
| CPK | · |

Abbreviations: ALT = alanine aminotransferase; AST = aspartate aminotransferase; CPK = creatine phosphokinase; GGT = gamma glutamyl transferase; Ig = immunoglobulin; INR = international normalized ratio; RBC = red blood cells; WBC = white blood cells.

- a Assayed by Lilly-designated laboratory.
- b Reflex/confirmation dependent on regulatory requirements and/or testing availability.

## **Attachment 4. Protocol JPBK ECOG Performance Status**

#### **ECOG Performance Status**

| <b>Activity Status</b> | Description |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but<br>ambulatory and able to carry out work of a light or<br>sedentary nature, e.g., light house work, office work |
| 2 | Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair |
| 5 | Dead. |

Source: Oken et al. 1982.
#### Attachment 5. Protocol JPBK RECIST Criteria 1.1

Response and progression will be evaluated in this study using the international criteria proposed by the New Response Evaluation Criteria in Solid Tumors (RECIST): Revised RECIST Guideline (version 1.1; Eisenhauer et al. 2009).

#### Measurability of Tumor at Baseline

Tumor lesions/lymph nodes will be categorized at baseline as measurable or nonmeasurable. Measurable disease is defined by the presence of at least 1 measurable lesion.

#### Measurable

Tumor lesions: Measured in at least 1 dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of:

- 10 mm by computed tomography (CT) or magnetic resonance imaging (MRI) scan (slice thickness ≤5 mm)
- 10 mm caliper measurement by clinical exam (non-measurable lesions if cannot be accurately measured with calipers)
- 20 mm by chest X-ray.

Malignant lymph nodes: To be considered pathologically enlarged and measurable, a lymph node must be  $\ge 15$  mm in short axis when assessed by CT scan (CT scan thickness recommended to be  $\le 5$  mm).

#### Nonmeasurable

All other lesions, including small lesions (longest diameter <10 mm or pathological lymph nodes with ≥10 to <15 mm short axis) as well as truly nonmeasurable lesions. Lesions considered truly non-measurable include: leptomeningeal disease, ascites, pleural/pericardial effusions, lymphangitis cutis/pulmonis, inflammatory breast disease, lymphangitis involvement of skin or lung, abdominal masses/abdominal organomegaly identified by physical exam that is not measureable by reproducible imaging techniques.

#### Special Considerations for Lesion Measurability

#### Bone lesions:

- Bone scan, PET scan or plain films are not considered adequate imaging techniques to measure bone lesions.
- Lytic bone lesions or mixed lytic-blastic lesions, with identifiable soft tissue components, that can be evaluated by cross sectional imaging techniques such as CT or MRI, can be considered measurable lesions if the soft tissue component meets the definition of measurability.
- Blastic bone lesions are non-measurable.

#### **Cystic lesions**:

- Simple cysts should not be considered as malignant lesions (neither measurable nor nonmeasurable)
- Cystic lesions thought to represent cystic metastases can be considered as measurable lesions, if they meet the definition of measurability. If noncystic lesions are presented in the same patients, these are preferred for selection as target lesions.

#### Lesions with Prior Local Treatment:

• Tumor lesions situated at a previously irradiated area, or in an area subjected to other loco-regional therapy, are non-measurable unless there has been demonstrated progression in the lesion.

#### **Baseline Documentation of Target and Non-Target Lesion**

#### **Target Lesions**

When more than 1 measurable lesion is present at baseline, all lesions up to a maximum of 5 lesions total (and a maximum of 2 lesions per organ) representative of all involved organs should be identified as target lesions and will be recorded and measured at baseline. Non-nodal Target lesions should be selected on the basis of their size (lesions with the longest diameter), be representative of all involved organs, and can be reproduced in repeated measurements.. Measurable lymph nodes are target lesions if they meet the criteria of a short axis of ≥15 mm by CT scan. All measurements are to be recorded in the case record form (CRF) in millimeters (or decimal fractions of centimeters [cm]).

#### Nontarget Lesions

All other lesions (or sites of disease) are identified as nontarget lesions (chosen based on their representativeness of involved organs and the ability to be reproduced in repeated measurements) and should be recorded at baseline. Measurement of these lesions are not required but should be followed as 'present,' 'absent,' or in rare cases 'unequivocal progression.' In addition, it is possible to record multiple nontarget lesions involving the same organ as a single item on the CRF (for example, multiple liver metastases recorded as 1 liver lesion).

Lymph nodes with short axis  $\geq 10$  mm but < 15 mm should be considered nontarget lesions. Nodes that have a short axis < 10 mm are considered nonpathological and are not recorded or followed.

#### **Specifications by Methods of Measurement**

All measurements should be recorded in metric notation, using a ruler or calipers if clinically assessed. All baseline evaluations should be performed as closely as possible to the beginning of treatment and never more than 4 weeks before the beginning of the treatment.

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during follow-up. Imaging-based evaluation is

should always be done rather than clinical examination unless the lesion(s) being followed cannot be imaged but are assessed by clinical exam.

An adequate volume of a suitable contrast agent should be given so that the metastases are demonstrated to best effect and a consistent method is used on subsequent examinations for any given patient. If prior to enrollment it is known a patient is not able to undergo CT scans with IV contrast due to allergy or renal insufficiency, the decision as to whether a non-contrast CT or MRI (with or without IV contrast) should be used to evaluate the patient at baseline and follow-up should be guided by the tumor type under investigation and the anatomic location of the disease.

Clinical Lesions: Clinical lesions will only be considered measurable when they are superficial and ≥10 mm diameter as assessed using calipers (for example, skin nodules). For the case of skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion is recommended. When lesions can be evaluated by both clinical exam and imaging, imaging evaluation should be undertaken since it is more objective and may be reviewed at the end of the study.

*Chest X-ray*: Chest CT is preferred over chest X-ray when progression is an important endpoint. Lesions on chest X-ray may be considered measurable if they are clearly defined and surrounded by aerated lung.

CT and MRI: CT scan is the best currently available and reproducible method to measure lesions selected for response assessment. Measurability of lesions on CT scan is based on the assumption that CT slice thickness is ≤5 mm. When CT scan have slice thickness >5 mm, the minimum size for a measurable lesion should be twice the slice thickness. MRI is also acceptable in certain situations (for example, for body scans). If there is concern about radiation exposure at CT, MRI may be used instead of CT in selected instances.

*Ultrasound:* Ultrasound should not be used to measure lesion size. Ultrasound examinations cannot be reproduced in their entirety for independent review at a later date and, because they are operator dependent, it cannot be guaranteed that the same technique and measurements will be taken from one assessment to the next. If new lesions are identified by ultrasound in the course of the study, confirmation by CT or MRI is advised.

*Endoscopy, Laparoscopy*: The utilization of these techniques for objective tumor evaluation is not advised. However, such techniques can be useful to confirm complete pathological response when biopsies are obtained or to determine relapse in trials where recurrence following complete response or surgical resection is an endpoint.

*Tumor Markers*: Tumor markers alone cannot be used to assess tumor response. If markers are initially above the upper normal limit, they must normalize for a patient to be considered in complete response (CR). Specific guidelines for both prostate-specific antigen (PSA) response (in recurrent prostate cancer) and CA-125 response (in recurrent ovarian cancer) have been published.

Cytology, Histology: These techniques can be used to differentiate between partial responses (PR) and complete response (CR) in rare cases if required by protocol (for example, residual lesions in tumor types such as germ cell tumors, where known residual benign tumors can remain). When effusions are known to be a potential adverse effect of treatment (for example, with certain taxane compounds or angiogenesis inhibitors), the cytological confirmation of the neoplastic origin of any effusion that appears or worsens during treatment can be considered if the measurable tumor has met criteria for response or SD in order to differentiate between response (or SD) and progressive disease (PD).

*Pet Scan (FDG-PET, PET CT)*: PET is not recommended for lesion assessment. If a new lesion is found by PET, another assessment must be done by CT, unless the PET CT is of diagnostic quality. If CT is done to confirm the results of the earlier PET scan, the date of progression must be reported as the earlier date of the PET scan.

*Bone Scan*: If lesions measured by bone scan are reported at baseline, it is necessary to repeat the bone scan when trying to identify a complete response (CR) or partial response (PR) in target disease or when progression in bone is suspected.

#### **Response Criteria**

#### **Evaluation of Target Lesions**

Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Tumor marker results must have normalized.

Partial Response (PR): At least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters.

*Progressive Disease (PD):* At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 or more new lesions is also considered progression.

For equivocal findings of progression (for example, very small and uncertain new lesions; cystic changes or necrosis in existing lesions), treatment may continue until the next scheduled assessment. If at the next scheduled assessment, progression is confirmed, the date of progression should be the earlier date when progression was suspected.

Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

*Not Evaluable:* When an incomplete radiologic assessment of target lesions is performed or there is a change in the method of measurement from baseline that impacts the ability to make a reliable evaluation of response.

#### **Evaluation of Nontarget Lesions**

*Complete Response:* Disappearance of all nontarget lesions and normalization of tumor marker level. All lymph nodes must be non-pathological or normal in size (<10mm short axis).

*Non-CR/ non-PD:* Persistence of 1 or more nontarget lesions and/or maintenance of tumor marker level above the normal limits.

*Progressive Disease:* Unequivocal progression of existing nontarget lesions. The appearance of 1 or more new lesions is also considered progression.

*Not Evaluable*: When a change in method of measurement from baseline occurs and impacts the ability to make a reliable evaluation of response.

#### **Evaluation of Best Overall Response**

The best overall response (BOR) is the best response recorded from the start of the study treatment until the earliest of objective progression or start of new anticancer therapy, taking into account any requirement for confirmation. The patient's best overall response assignment will depend on the findings of both target and nontarget disease and will also take into consideration the appearance of new lesions. The BOR will be calculated via an algorithm using the assessment responses provided by the investigator over the course of the trial.

#### Time Point Response

It is assumed that at each protocol-specified time point, a response assessment occurs. (When no imaging/measurement is done at all at a particular time point, the patient is not evaluable (NE) at that time point.) Table 1 provides a summary of the overall response status calculation at each time point for patients who have *measurable disease* at baseline.

Table 1. Time Point Response: Patients with Target (± Nontarget) Disease

| <b>Target Lesions</b> | Non-Target Lesions | <b>New Lesions</b> | Overall Response |
|---|---|---|---|
| CR | CR | No | CR |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not all evaluated | No | PR |
| SD | Non-PD or not all evaluated | No | SD |
| Not all evaluated | Non-PD | No | NE |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |

Abbreviations: CR = complete response; PR = partial response; SD = stable disease.; PD = progressive disease; NE = inevaluable.

Table 2 is to be used when patients have *nonmeasurable* disease only.

| rabio 2 | | |
|-------------------|-------------|----------------------------|
| Nontarget Lesions | New Lesions | Overall Response |
| CR | No | CR |
| Non-CR/non-PD | No | Non-CR/non-PD <sup>a</sup> |
| Not all evaluated | No | NE |
| Unequivocal PD | Yes or No | PD |
| Any | Yes | PD |

Table 2. Time Point Response: Patients with Nontarget Disease Only

Abbreviations: CR = complete response; PD = progressive disease; NE = inevaluable.

#### Frequency of Tumor Re-Evaluation

A baseline tumor evaluation must be performed within 4 weeks before patient begins study treatment. Frequency of tumor re-evaluation while on and adapted to treatment should be protocol-specific and adapted to the type and schedule of treatment. In the context of Phase 2 studies where the beneficial effect therapy is not known, follow-up every 6-8 weeks is reasonable. Normally, all target and non-target sites are evaluated at each assessment using the same method. However, bone scans may need to be repeated only when CR is identified in target disease or when progression in bone is suspected.

#### **Confirmatory Measurement/Duration of Response**

#### Confirmation:

The main goal of confirmation of objective response in clinical trials is to avoid overestimating the response rate observed. The confirmation of response is particularly important in *nonrandomized trials* where response (CR/PR) is the primary end point. In this setting, to be assigned a status of PR/CR, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 4 weeks after the criteria for response are first met. To confirm a response of CR, a full assessment of all target and nontarget lesions that were present at baseline must occur, including those measured by bone scan. To confirm a PR or SD, a full assessment of target lesions that were present at baseline must occur; assessment of nontargets is not required.

However, in *randomized trial* (Phase 2 or 3) or studies where SD or progression is the primary endpoints, confirmation of response is not required. But, elimination of the requirement may increase the importance of central review to protect against bias, in particular of studies which are not blinded.

In the case of SD, follow-up measurements must have met the SD criteria at least once after start of treatment at a minimum interval not less than 6 weeks measured from first dose.

#### Duration of Overall Response

The duration of overall response is measured from the time measurement criteria are first met for CR or PR (whichever is first recorded) until the first date that disease is recurrent or objective progression is observed (taking as reference for PD the smallest measurements recorded on study).

<sup>&</sup>lt;sup>a</sup> non-CR/non-PD is preferred over SD for nontarget disease.

The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented.

#### Duration of Stable Disease

Stable disease is measured from the start of the treatment (in randomized trials, from date of randomization) until the criteria for objective progression are met, taking as reference the smallest sum on study (if the baseline sum is the smallest, that is the reference for calculation of PD).

#### **Independent Review of Response and Progression**

When objective response (CR + PR) is the primary end point, and when key drug development decisions are based on the observation of a minimum number of responders, it is recommended that all claimed responses be reviewed by an expert(s) independent of the study. If the study is a randomized trial, ideally reviewers should be blinded to treatment assignment.

### **Attachment 6. Protocol JPBK Sampling Summary**

This table summarizes the maximum number of samples (venipunctures, biopsies), volumes for all sampling, and tests (study qualification, health monitoring, drug concentration, pharmacodynamics/tailoring biomarkers) during the study. The summary below provides estimates. More samples could be required in the case of retests, additional health monitoring (if needed), or for patients continuing treatment beyond the protocol-specified number of cycles in the study. Fewer samples may actually be taken (for example, patients who discontinue from the study).

Protocol I3Y-MC-JPBK Sampling Summary<sup>a</sup>

| | Sample | Maximum Amount | Maximum Number | Maximum |
|---|---|---|---|---|
| Purpose | Type | per Sample | Samples | Total Amount |
| Study qualification <sup>b</sup> | Blood | 6 mL | 1 | 6 mL |
| KRAS mutant status <sup>b</sup> | FFPE tumor<br>tissue slides<br>or block | FFPE tumor tissue<br>slides<br>OR<br>FFPE tumor tissue<br>block | 8 slides OR 1 tumor tissue block | FFPE tumor<br>tissue slides or<br>block |
| Tissue for biomarker research | FFPE tumor<br>tissue slides<br>or block | FFPE tumor tissue<br>slides<br>OR<br>FFPE tumor tissue<br>block | 20 slides 5 micron<br>thickness<br>OR<br>1 tumor tissue block | FFPE tumor<br>tissue slides or<br>block |
| Health monitoring <sup>a</sup> | Blood for chemistry | 3 mL | 13 | 39 mL |
| | Blood for<br>Hematology | 3 mL | 13 | 39 mL |
| Drug concentration | Blood | 2 mL | 5 | 10 mL |
| Pharmacodynamics and/or other biomarkers | Blood | 10 mL | 2 | 20 mL |
| Stored sample for pharmacogenetic evaluations | Blood | 6 mL | 1 | 6 mL |
| Hepatic monitoring <sup>c</sup> | Blood | 3 - 30 mL | - | - |
| Total: Blood | | | | 120 mL |

Abbreviation: FFPE = formalin-fixed paraffin-embedded.

a Covers 12 cycles and Visit 801.

b This sample is required for initial qualification. The remaining samples are for those patients enrolled in the study.

c Based on laboratory safety values, unscheduled hepatic monitoring testing may be performed as part of patient follow-up, in consultation with the designated medical monitor.

# Attachment 7. Protocol JPBK Pharmacokinetic Sampling Schedule

#### **Pharmacokinetic Sampling Schedule**

| PK Sample<br>Number | Cycle (C)<br>and Day (D) | Dosing of<br>LY2835219 | Sampling Time for PK from Blood <sup>a</sup> |
|---|---|---|---|
| 1 | C1D1 | $X^{b}$ | 4-6 hrs after LY2835219 dose |
| 2 | C2D1 | X <sup>c</sup> | At least 4 hrs after taking LY2835219 dose at home (that is, upon arrival at site) |
| 3 | C2D1 | | At least $7 \pm 0.5$ hrs after taking LY2835219 dose at home (that is, $3 \pm 0.5$ hrs after arrival at site) |
| 4 | C3D1 | X | Prior to LY2835219 dose |
| 5 | C3D1 | | $3 \pm 0.5$ hrs after LY2835219 dose |

Abbreviations: C = Cycle; D = Day; ECG = electrocardiogram; hr = hour; LY = LY2835219; PK = pharmacokinetic; Q12H = every 12 hours.

- <sup>a</sup> Samples of approximately 2 mL of whole blood will be drawn, for measurement of LY2835219 and its metabolites concentrations in plasma.
- b On Cycle 1 Day 1 only, patients should take 1 single dose of LY2835219 and initiate chronic Q12H dosing on Cycle 1 Day 2.
- <sup>c</sup> On Cycle 2 Day 1 only, patient should take LY2835219 dose at home at approximately 4 hours before arrival at site. The time of LY2835219 dose intake must be recorded that day.

## Attachment 8. Protocol JPBK Inducers and Strong Inhibitors of CYP3A4 or Substrates of CYP2B6

The information in this attachment is provided for guidance to investigators and does not preclude the use of these medications if clinically indicated.

#### **Inducers of CYP3A4**

Carbamazepine

Dexamethasone<sup>a</sup>

Phenobarbital/phenobarbitone

Phenytoin

Rifapentine

Rifampin

Rifabutin

St. John's wort

#### Strong inhibitors of CYP3A4

All HIV protease inhibitors

Clarithromycin

Itraconazole

Ketoconazole

Nefazodone

a Important note: All patients may receive supportive therapy with dexamethasone, preferably ≤7 days, if clinically indicated. A patient who develops brain metastases may receive acute or chronic therapy with dexamethasone if clinically indicated. Development of brain metastases is considered progressive disease and the patient should discontinue study treatment.

#### **Substrates of CYP2B6**

Alfentanil

**Bupropion** 

cyclophosphamide

Efavirenz

Ifosfamid

methadone

Nevirapine

Propofol

Sertraline

sorafenib

tamoxifen

Valproic acid

CCI

Approver: PPD

Approval Date & Time: 13-May-2014 12:22:23 GMT Signature meaning: Approved

Approver: PPD

Approval Date & Time: 13-May-2014 13:21:14 GMT Signature meaning: Approved

Leo Document ID = 01295e39-6509-458f-a6e1-173358aad1f8

Approver: PPD

Approval Date & Time: 10-Jul-2018 09:10:11 GMT Signature meaning: Approved

Leo Document ID = 01295e39-6509-458f-a6e1-173358aad1f8

Approver: PPD

Approval Date & Time: 11-Jul-2018 20:06:14 GMT Signature meaning: Approved

Leo Document ID = 26b45807-4b57-4011-b552-84b053823872

Approver: PPD

Approval Date & Time: 23-Aug-2018 14:44:33 GMT Signature meaning: Approved